# An open-label, multicentre study to evaluate pharmacokinetics, safety and efficacy of zamicastat as adjunctive therapy in pulmonary arterial hypertension (PAH)

Sponsor Project Code: BIA-51058-201 Scope Project Code: 0223BI26.MPB

## STATISTICAL ANALYSIS PLAN

Sponsor: Bial - Portela & Ca, S.A.

À Av. da Siderurgia Nacional

4745-457 Coronado (S. Romão e S. Mamede), Portugal

Phone: +351 229866100 Fax: +351 229866192

Author: Lukas Pukys

Statistician

Scope International AG

Kalvariju 300

LT-08318 Vilnius, Lithuania

E-mail: lpukys@scope-international.com

Phone: +370 5 2361 833 Fax: +370 5 2388 533

**Version:** Final 1.0 (22-MAR-2022)

The information provided in this document is strictly confidential. No part of this document may be reproduced, transmitted or copied in any form nor its contents disclosed to the third parties without prior written consent of Bial - Portela & Ca, S.A. or a nominated representative.

#### **DOCUMENT REVISION HISTORY**

Version Draft 0.1 (09-JUL-2021): Document was created.

Version Draft 0.2 (07-SEP-2021): Document updated after sponsor's review. Notable changes:

- Added table 15.2.5.1 (section 5.5.5)
- Removed the original SF-6D score from analysis (section 5.5.6)
- Added figures 15.2.1 and 15.2.2 (section 5.5.6)
- Added the definition of TEAEs leading to down-titration and table 15.3.1.7 (section 5.6.1)
- Added table 15.3.5.4.2 (section 5.6.5)

Version Draft 0.3 (24-NOV-2021): Document updated after sponsor's review. Notable changes:

- Added specification that the definition of PAH medications will be reviewed during the DRM (section 5.3)
- Updated the range of nominal compliance to 90%-110% (section 5.4.2)
- Added within-visit shift table for ECG abnormalities (section 5.6.5)

Version Draft 0.4 (06-JAN-2022): Document updated after the Data Review meeting and the sponsor's review. Notable changes:

- Changed definition of FAS to only include patients with non-missing efficacy assessments at MPV3 (Section 3.1)
- Added definition of mFAS (Section 3.1). Efficacy analyses will be performed for both the FAS and MFAS (Section 5.5).
- Added definitions for TAPSE subgroups (Section 3.2). TAPSE subgroup analyses will be performed for selected efficacy parameters (Sections 5.5.1, 5.5.2, 5.5.4)
- Safety data will no longer be summarised at derived visit V3. Actual visits will be used (Section 4.4)
- Added definition of PAH-approved medications and corresponding tables (Section 5.3)
- Right heart catheterisation clinical significance assessments will not be used in statistical analysis (Section 5.5.1)
- Added specification that in case the distance covered during both 6MWT attempts is equal, the first attempt will be considered as baseline (Section 5.5.2)
- Changed unit for biomarket NT-proBNP from pg/mL to ng/L (Section 5.5.3)
- Added specification for interpreting normal, NCS abnormal, and CS abnormal findings for arterial blood gas analysis (Section 5.6.3) and ECG (Section 5.6.5)

Version Draft 0.5 (08-FEB-2022): Document updated after sponsor's review. Notable changes:

• Added the coefficient of variance to standard summary statistics (Section 4.1)

Version Draft 0.6 (17-MAR-2022): Document updated after sponsor's review. Notable changes:

• Amended the definition of PAH-approved medications to include diuretics (Sections 3.1, 5.3) Version Final 1.0 (22-MAR-2022): Document finalised.

I-DM-011SAP 

## TABLE OF CONTENTS

| L | JST OF ABBREVIATIONS AND KEY TERMS | 5 |
|----|---------------------------------------------------------|----|
| II | NTRODUCTION | 7 |
| 1 | FLOW CHART AND VISIT SCHEDULE | 8 |
| | 1.1 FLOW CHART | 8 |
| | 1.2 SCHEDULE OF STUDY PROCEDURES | 9 |
| 2 | OBJECTIVES AND DESIGN | 12 |
| | 2.1 Study Objectives | 12 |
| | 2.1.1 Primary Objective | |
| | 2.1.2 Secondary Objectives | |
| | 2.2 Study Endpoints | |
| | 2.2.1 Primary Endpoint | |
| | 2.2.2 Secondary Endpoints | |
| | 2.2.2.1 Safety Endpoints | |
| | 2.2.2.3 Pharmacokinetic Endpoints | |
| | 2.2.2.4 Pharmacodynamic Endpoints | |
| | 2.3 OVERALL STUDY DESIGN | |
| | 2.4 RANDOMISATION | |
| | 2.5 Treatment | |
| | 2.6 SAMPLE SIZE | 15 |
| | 2.7 Blinding | 16 |
| 3 | ANALYSIS SETS AND SUBGROUPS | 17 |
| | 3.1 Analysis Sets | 17 |
| | 3.2 SUBGROUP ANALYSIS | |
| 4 | GENERAL DEFINITIONS AND NAMING CONVENTIONS | 18 |
| | 4.1 GENERAL METHODOLOGY AND PRESENTATION OF THE RESULTS | 18 |
| | 4.2 STATISTICAL OUTPUT LAYOUT | |
| | 4.3 Dose Group Names and Labels | |
| | 4.4 VISIT NAMES AND LABELS | |
| | 4.5 DAY NUMBERING | |
| | 4.6 STUDY PERIODS | |
| | 4.7 BASELINE VALUE | |
| | 4.9 CODING SYSTEMS AND CONVENTIONS | |
| | 4.9.1 Coding of adverse events and medical history | |
| | 4.9.2 Coding of medications | |
| | 4.10 HANDLING OF MISSING DATA | |
| 5 | , | |
| | METHODOLOGY | 22 |
| | 5.1 PATIENT DISPOSITION | |
| | 5.1.1 Disposition and Withdrawals | |
| | 5.1.2 Protocol Deviations | |
| | 5.1.3 Inclusion/Exclusion | |
| | 5.2.1 Demographics | |
| | 5.2.1 Demographics | |
| | 5.2.3 Medical History | |
| | 5.3 PRIOR AND CONCOMITANT MEDICATIONS | |

| 5.4 EXPOSURE TO IMP AND COMPLIANCE | 27 |
|--------------------------------------------------------------------|----|
| 5.4.1 Exposure to IMP | |
| 5.4.2 Compliance | |
| 5.5 ANALYSIS OF EFFICACY ENDPOINTS | 29 |
| 5.5.1 Right Heart Catheterisation | |
| 5.5.2 6-Min Walk Test (6-MWT) | |
| 5.5.3 Biomarker | |
| 5.5.4 Echocardiography | |
| 5.5.5 New York Heart Association/Word Health Organisation Function | |
| (NYHA/WHO)5.5.6 Ouality of Life (SF-36v2) | |
| 5.5.6 Quality of Life (SF-36v2) | |
| 5.6.1 Adverse Events | |
| 5.6.2 Clinical Laboratory Evaluation | |
| 5.6.3 Arterial Blood Gas Analysis | |
| 5.6.4 Vital Signs | |
| 5.6.5 12-Lead Electrocardiogram (ECG) Data | |
| 5.6.6 Physical Examination Findings | |
| 5.6.7 Number of Digital Scars | 42 |
| 5.6.8 Modified Rodnan Skin Score (mRSS) | 42 |
| 6 DATA REVIEW | 44 |
| 7 INTERIM ANALYSIS | 48 |
| 8 CHANGES TO THE ANALYSIS AS LAID DOWN IN THE PROTOCOL AND | ` |
| AMENDMENTS | |
| 9 REFERENCES | 50 |
| 10 APPENDICES | 51 |
| 10.1 Tables | 51 |
| 10.2 Listings | |
| 10.3 Figures | |
| SIGNATURES | 59 |

## LIST OF ABBREVIATIONS AND KEY TERMS

| Abbreviations | Description of abbreviations |
|---|---|
| 6-MWT | 6-minute walk test |
| $\lambda_{\rm z}$ | Terminal rate constant |
| AE | Adverse event |
| ALT | Alanine transaminase |
| AST | Aspartate transaminase |
| AUC | Area under the curve |
| AUEC | Area under the effect-time curve |
| CI | Cardiac index |
| CL/f | Apparent total clearance |
| $C_{max}$ | Maximum plasma concentration |
| $C_{\min}$ | Minimum plasma concentration |
| СО | Cardiac output |
| CPK | Creatine phosphokinase |
| CS | Clinically significant |
| CV | Coefficient of variation |
| DßH | Dopamine β-hydroxylase |
| DBP | Diastolic blood pressure |
| DPG | Diastolic pressure gradient |
| DR(M) | Data review (meeting) |
| DSMB | Data safety monitoring board |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| EDV | Early discontinuation visit |
| $E_{\text{max}}$ | Maximum observed effect on DβH activity |
| ES | Enrolled set |
| FAS | Full analysis set |
| GGT | Gamma-glutamyl transferase |
| HbA1c | Haemoglobin A1c |
| HCG | Human chorionic gonadotropin |
| HTD | Highest tolerated dose |
| ICF | Informed consent form |
| IMP | Investigational medicinal product |
| LDH | Lactate dehydrogenase |
| LLOQ | Lower limit of quantification |
| LPLV | Last patient's last visit |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mPAP | Mean pulmonary artery pressure |
| mRSS | Modified Rodnan skin score |
| NCS | Not clinically significant |
| NT-proBNP | N-terminal pro brain natriuretic peptide |
| NYHA/WHO | New York Heart Association/Word Health Organisation |
| PAC | Pulmonary arterial compliance |
| PAH | Pulmonary arterial hypertension |
| PAPs | Pulmonary artery pressure systolic |
| PAPd | Pulmonary artery pressure diastolic |
| PAWP | Pulmonary artery wedge pressure |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| PKS | Pharmacokinetic analysis set |

I-DM-011SAP 

| PT | Preferred term |
|---|---|
| PVR | Pulmonary vascular resistance |
| RAP | Right atrial pressure |
| RBC | Red blood cell count |
| RHC | Right heart catheterisation |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS | Statistical Analysis System |
| SBP | Systolic blood pressure |
| SF-36 | Short Form - 36 |
| $S_vO_2$ | Mixed venous oxygen saturation |
| SOC | System organ class |
| SS | Safety set |
| SVR | Systemic ventricular resistance |
| t <sub>1/2</sub> | Terminal half-life |
| TAPSE | Tricuspid annular plane systolic excursion |
| TEAE | Treatment emergent adverse event |
| $T_{Emax}$ | Time to occurrence of $E_{max}$ |
| t <sub>max</sub> | Time until C <sub>max</sub> |
| TPG | Transpulmonary pressure gradient |
| UV | Unscheduled visit |
| V | Visit |
| V <sub>z</sub> /f | Apparent volume of distribution |
| WBC | White blood cell count |
| WHO World Health Organization | |
| ZMC | Zamicastat |

I-DM-011SAP Effective date: 15.09.2020 

#### **INTRODUCTION**

This statistical analysis plan (SAP) contains a more technical and detailed elaboration of the principal features of the statistical analyses as described in the clinical study protocol versions:

| Document, Version | Date |
|------------------------|-------------|
| Protocol, Final 1.0 | 22-JUN-2018 |
| Protocol, Final 2.0 | 18-JUN-2019 |
| Protocol, Final 2.0 UK | 08-JUL-2019 |
| Protocol, Final 2.0 DE | 23-SEP-2019 |
| Protocol, Final 3.0 | 12-MAY-2020 |

This SAP is written assuming the latest version (**Final 3.0**, 12-MAY-2020). Relevant differences between the protocol versions will be listed in the corresponding subsections of the SAP.

This SAP includes detailed procedures for executing the statistical analysis of the secondary safety, tolerability and efficacy variables and other data, and it is structured according to different data types. The SAP is finalised and signed-off before analysis begins in an open-label study. This SAP supersedes statistical considerations previously defined in the clinical study protocol. Analysis of the primary endpoint (pharmacokinetics (PK)) as well as secondary PK and pharmacodynamics (PD) endpoints is covered in a separate reporting and analysis plan prepared by Quotient Sciences Ltd (Appendix 4).

All analysis data sets and statistical output related to the secondary safety, tolerability and efficacy endpoints will be produced by the statistics department of Scope International AG using SAS® for Windows (SAS Institute Inc., Cary, NC, USA) [1] version 9.4 or higher. The actual version used will be documented in the Validation Plan for Statistical Programming.

I-DM-011SAP 

#### 1 FLOW CHART AND VISIT SCHEDULE

#### 1.1 Flow Chart



I-DM-011SAP Effective date: 15.09.2020

## 1.2 Schedule of Study Procedures

| | Screening | | Dose finding pe | eriod | 42-days | Maintenance | period | Foll | ow-up |
|---|---|---|---|---|---|---|---|---|---|
| Visit no. | V1 | A1 <sup>2</sup> | A2/B2/C2/D2 | A3/B3/C3/D3 <sup>5</sup> | MPV1 <sup>5</sup> | MPV2 <sup>5</sup> | MPV3 <sup>2,5</sup> /<br>EDV <sup>1</sup> | Follow-up<br>down-<br>titration <sup>7</sup> | FU <sup>17</sup> |
| | Day -12 to -5 | Day 1 | 8 days ±2 after<br>A1/A3/B3/C3 | 14 days ±2 after<br>A1/A3/B3/C3 | 13 days ±2<br>after<br>D3/down-<br>titration <sup>19</sup> | 27 days ±2<br>after D3/<br>down-<br>titration <sup>19</sup> | 41 days ±2<br>after D3/<br>down-<br>titration <sup>19</sup> | 14 days ±2<br>after<br>MPV3/EDV | 14 days ±2<br>after last IMP<br>intake |
| on-site visit ⊗ /<br>telephone contact <b>*</b> | 8 | $\otimes$ | <b>~</b> | 8 | 8 | 8 | 8 | <b>~</b> | 8 |
| Initiation procedures | | | | | | | | | |
| Informed consent | • | | | | | | | | |
| Demographics | • | | | | | | | | |
| Height | • | | | | | | | | |
| Weight | • | | | | | | • | | |
| Medical history | • | | | | | | | | |
| Prior medication | • | | | | | | | | |
| Concomitant medication | • | • | • | • | • | • | • | • | • |
| WHO functional class | • | | | | | | • | | |
| Inclusion/exclusion criteria | • | • | | | | | | | |
| Medication | | | | | | | | | |
| First IMP administration | | • | | | | | | | |
| Dose increase | | | | •3 | | | | | |
| Dispense IMP | | • | | • | • | • | ●7 | | |
| IMP accountability | | | | • | • | • | • | | ●7 |
| Pharmacokinetics/<br>Pharmacodynamics | | | | | | | | | |
| Blood withdrawal (24h profile) | | ●4 | | | | | ●4,8 | | |
| Blood withdrawal (trough level) | | | | ●14 | ●14 | ●14 | | | |
| Blood withdrawal (DβH activity) | | •4 | | ●14 | ●14 | ●14 | ●4,8 | | |
| Urinalysis (dopamine and norepinephrine levels, 24h urine collection) <sup>15</sup> | | • | | • | | | •8 | | |

I-DM-011SAP

| | Screening | | Dose finding pe | eriod | 42-days | Maintenance | period | Foll | ow-up |
|---|---|---|---|---|---|---|---|---|---|
| Visit no. | V1 | A1 <sup>2</sup> | A2/B2/C2/D2 | A3/B3/C3/D3 <sup>5</sup> | MPV1 <sup>5</sup> | MPV2 <sup>5</sup> | MPV3 <sup>2,5</sup> /<br>EDV <sup>1</sup> | Follow-up<br>down-<br>titration <sup>7</sup> | FU <sup>17</sup> |
| | Day -12 to -5 | Day 1 | 8 days ±2 after<br>A1/A3/B3/C3 | 14 days ±2 after<br>A1/A3/B3/C3 | 13 days ±2<br>after<br>D3/down-<br>titration <sup>19</sup> | 27 days ±2<br>after D3/<br>down-<br>titration <sup>19</sup> | 41 days ±2<br>after D3/<br>down-<br>titration <sup>19</sup> | 14 days ±2<br>after<br>MPV3/EDV | 14 days ±2<br>after last IMP<br>intake |
| on-site visit ⊗ /<br>telephone contact ☎ | 8 | $\otimes$ | <b>~</b> | 8 | 8 | 8 | 8 | <b>~</b> | 8 |
| Safety | | | | | | | | | |
| Adverse events | • | • | • | • | • | • | • | • | • |
| Vital signs <sup>11</sup> (blood pressure, heart rate, tympanic body temperature) | • | <b>●</b> 12 | | • | • | • | ●12 | | • |
| Blood withdrawal (haematology, biochemistry and coagulation) | • | | | • | • | | • | | • |
| Urinalysis | • | | | • | • | | • | | • |
| Physical examination | • | | | • | • | • | • | | |
| 12-lead electrocardiogram | • | ●18 | | • | • | • | ●18 | | • |
| Number of digital scars <sup>10</sup> | • | | | • | • | • | • | | |
| Modified Rodnan Skin Score <sup>10</sup> | • | | | | | | • | | |
| Blood pregnancy test <sup>6</sup> | • | | | | | | | | |
| Urine pregnancy test <sup>6</sup> | | • | | • | • | • | • | | • |
| Arterial blood gas analysis 16,21 | | • | | | | | •8 | | |
| Efficacy | | | | | | | | | |
| SF-36v2 | • | | | | | | •8 | | |
| 6-min walk test/Borg dyspnoea score | ●13 | | | | | | ●8,20 | | |
| Echocardiography | • | | | | | | •8 | - | |
| Right heart catheterisation 16,22 | | • | | | | | •8 | - | |
| Blood withdrawal biomarker | • | <u></u> | | | | | ●8 | | |

<sup>1.</sup> EDV = early discontinuation visit. An EDV has to be performed within 10 days of early discontinuation. Additionally, patients who will not participate in the extension study will be contacted by phone at the time of last patient's last visit (LPLV) to document their vital status.

I-DM-011SAP Effective date: 15.09.2020

<sup>2.</sup> Patients will be hospitalised for 24 hours.

- 3. The dose will be increased if the previous dose was considered safe by the investigator according to safety criteria (at A3, B3 and C3).
- 4. Blood samples for PK and PD to be taken prior to IMP intake as well as 1, 2, 4, 8, 16 and 24 hours after IMP intake (but still prior to next IMP intake).
- 5. The patient has to be advised not to take the IMP at home on the day of A3, B3, C3, D3, MPV1, MPV2 and MPV3.
- 6. Only in women of childbearing potential.
- 7. Only applicable in patients taking 150 mg or 200 mg zamicastat and who will not participate in the extension study. In case a patient will discontinue the study early due to the occurrence of an AE, down-titration is not mandatory, but at the investigator's discretion.
- 8. Not applicable at EDV.
- 9. Visits during the Dose-finding period:

Dose A (50 mg zamicastat): visits A1, A2 and A3

Dose B (100 mg zamicastat): visits B2 and B3. These visits will only be performed if the patient was up-titrated to 100 mg zamicastat at A3.

Dose C (150 mg zamicastat): C2 and C3. These visits will only be performed if the patient was up-titrated to 150 mg zamicastat at B3.

Dose D (200 mg zamicastat): D2 and D3. These visits will only be performed if the patient was up-titrated to 200 mg zamicastat at C3.

If the patient's next dose will not be tolerated, the patient will be asked to come to an unscheduled visit (UV) and he/she will be down-titrated to his/her previous dose. 10. In scleroderma patients only.

- 11. Blood pressure and heart rate will be measured in supine position (two measurements) and afterwards in standing position (one measurement).
- 12. At A1 and MPV3 blood pressure and heart rate (two measurements in supine and one measurement in standing position) will be measured before IMP intake as well as 4, 8 and 24 hours after IMP intake.
- 13. Two baseline tests, separated by an interval of at least 30 minutes.
- 14. Blood samples will be taken prior to IMP intake.
- 15. 24-hour urine collection will start on the day before the respective visit.
- 16. Right heart catheterisation and arterial blood gas analysis have to be performed before IMP intake.
- 17. Applicable in all patients who will not participate in the extension study as well as in patients who discontinued early.
- 18. At A1 and MPV3 triplicate ECGs recordings will be performed before IMP intake, 4 and 8 hours after IMP intake. At EDV only one ECG recording will be performed.
- 19. Down-titration can be performed at a scheduled visit or an unscheduled visit (on-site visit or telephone contact) during the dose finding period.
- 20. 6-MWT has to be performed after arterial blood gas analysis but before right heart catheterisation and IMP intake.
- 21. Arterial blood gas analysis has to be performed before right heart catheterisation.
- 22. Right heart catheterisation will only be performed if no results which were measured at the study site from within 90 days before V1 are available.

I-DM-011SAP 

#### 2 OBJECTIVES AND DESIGN

## 2.1 Study Objectives

## 2.1.1 Primary Objective

The primary objective of this study is to evaluate the PK profile of different zamicastat doses in pulmonary arterial hypertension (PAH) patients to find the most promising therapeutic dosage range for the treatment of PAH disease. This SAP does not cover the analysis of the primary objective.

## 2.1.2 Secondary Objectives

The secondary objectives of this study are:

- 1. To assess further PK parameters including apparent total clearance, terminal half-life and apparent volume of distribution \*
- 2. To assess the safety and tolerability of different zamicastat doses
- 3. To investigate the effect of different zamicastat doses on plasma dopamine β hydroxylase (DβH) activity\*
- 4. To investigate the effect of different zamicastat doses on urinary catecholamine levels (norepinephrine and dopamine)\*
- 5. To investigate the change in pulmonary haemodynamic parameters
- 6. To investigate the change in the 6-minute walk test (6-MWT)
- 7. To investigate the change in biomarkers
- 8. To investigate the change in cardiac structure and contractibility, assessed by echocardiography
- 9. To investigate the change in quality of life, assessed by SF-36v2
  - \* Covered in a reporting and analysis plan prepared by Quotient Sciences Ltd. (Appendix 4).

## 2.2 Study Endpoints

## 2.2.1 Primary Endpoint

The following PK parameters (24-hour profile) for zamicastat and its metabolites will be derived after a single dose of 50 mg zamicastat at visit A1 (Day 1):

- 1. Area under the curve 0-24 h (AUC<sub>0-24h</sub>)
- 2. Maximum plasma concentration (C<sub>max</sub>)
- 3. Time until  $C_{max}$  ( $t_{max}$ )

The following PK parameter (24-hour profile) for zamicastat and its metabolites will be derived at steady-state at the individual HTD and will be taken at visit MPV3:

- 4. Area under the curve 0-24 h (AUC<sub>0-24h,SS</sub>)
- 5. Maximum plasma concentration (C<sub>max.SS</sub>)
- 6. Time until  $C_{\text{max,SS}}(t_{\text{max,SS}})$
- 7. Minimum plasma concentration at the end of the dosing interval (C<sub>min.SS</sub>)

The following PK parameter (trough level) will be derived for each dose at steady-state (visits A3, B3, C3, D3, MPV1, MPV2, MPV3).

8. Minimum plasma concentration at the end of the dosing interval (C<sub>min,SS</sub>)

I-DM-011SAP 

The analysis of PK parameters is covered in a reporting and analysis plan prepared by Quotient Sciences Ltd. (Appendix 4).

## 2.2.2 Secondary Endpoints

## 2.2.2.1 Safety Endpoints

The safety endpoints of this study are:

- Adverse events
- 2. Clinically relevant changes in laboratory parameters (haematology, biochemistry, coagulation, urinalysis, arterial blood gas analysis)
- 3. Clinically relevant changes in vital signs
- 4. Clinically relevant changes in physical examination
- 5. Clinically relevant changes in ECG
- 6. Number of digital scars (only in patients with scleroderma)
- 7. Skin score (only in patients with scleroderma)

## 2.2.2.2 Efficacy Endpoints

The secondary efficacy endpoints of this study are the change from baseline to visit MPV3 in:

- 8. Pulmonary vascular resistance (PVR), right atrial pressure (RAP), mean pulmonary artery pressure (mPAP), cardiac index (CI) and mixed venous oxygen saturation (S<sub>v</sub>O<sub>2</sub>). Further haemodynamic parameters may also be calculated if considered appropriate.
- 9. 6-MWT, including Borg dyspnoea score
- 10. Biomarker (NT-proBNP)
- 11. Echocardiogram parameters:
  - Tricuspid regurgitation, classified as absent, mild, moderate or severe
  - Right ventricular contractibility, measured via tricuspid annular plane systolic excursion (TAPSE)
  - Pericardial effusion, classified as absent, traces or present
  - Right atrial area (end-systolic), right ventricular end-diastolic area
- 12. WHO functional class
- 13. Quality of life (SF-36v2)

## 2.2.2.3 Pharmacokinetic Endpoints

- 14. Apparent total clearance (CL/f)
- 15. Terminal half-life  $(t_{1/2})$
- 16. Apparent volume of distribution (Vz/f)

The analysis of PK parameters is covered in a reporting and analysis plan prepared by Quotient Sciences Ltd. (Appendix 4).

I-DM-011SAP 

#### 2.2.2.4 Pharmacodynamic Endpoints

- 17. Percent inhibition in plasma DβH activity (i.e. % change from baseline of DβH activity) on visits A3/B3/C3/D3, MPV1 and MPV2 (trough samples) and to visits A1 and MPV3 (24-hour profiles)
- 18. Maximal and minimal observed effect on D $\beta$ H activity and time to occurrence of  $E_{max}$  ( $T_{Emax}$ ) and  $E_{min}$  ( $T_{Emin}$ ) on visit A1 (Day 1) and MPV3
- 19. Area under the effect-time curve (AUEC24) for % DβH inhibition on visit A1 (Day 1) and MPV3
- 20. Change from baseline 24-hour urinary catecholamine levels (norepinephrine and dopamine) on visits A3/B3/C3/D3 and MPV3.

The analysis of pharmacodynamic parameters is covered in a reporting and analysis plan prepared by Quotient Sciences Ltd. (Appendix 4).

## 2.3 Overall Study Design

This is an open-label, multi-centre study in patients with PAH who are currently on stable treatment with at least one PAH medication. It is planned to evaluate the PK profile (24-hour profile and trough levels) and the safety, tolerability and efficacy of four different zamicastat doses. Each patient will start treatment with the lowest dose (50 mg zamicastat once daily) and the dose will be up-titrated to the individual **highest tolerated dose** (HTD) i.e. up to 200 mg zamicastat once daily.

A data safety monitoring board (DSMB) will periodically review the safety data and will issue a recommendation if the doses can be used as planned.

This study will consist of:

- A screening period, 5 to 12 days: visit V1
- Up to four dose finding periods, 14 days each:

o Dose A: visits A1, A2 and A3 o Dose B: visits B2 and B3 o Dose C: visits C2 and C3 o Dose D: visits D2 and D3

- Maintenance period, 42 days: visits MPV1, MPV2 and MPV3
- <u>Follow-up period</u>:
  - o Visit FU (down-titration): 14 days after MPV3 (only for patients taking 150 mg or 200 mg zamicastat who will not participate in the extension study)
  - o Visit FU: 14 days after last IMP intake

After confirmed eligibility, patients will initiate treatment with Dose A (50 mg zamicastat once daily) at visit A1 and will be treated with this dose level for 14 days. If Dose A was considered safe by the investigator, the patient will be up-titrated to Dose B (100 mg zamicastat once daily) at visit A3 and the patient will continue with this dosage for 14 days. Patients not tolerating Dose A have to be withdrawn from the study.

After a positive safety evaluation at visit B3, the patient will be up-titrated to Dose C (150 mg zamicastat once daily) and the patient will continue on this dose level for a further 14 days. If Dose C was tolerated by the patient, he/she will be up-titrated at visit C3 to Dose D (200 mg zamicastat once daily) where the patient will remain for 56 days (14 days dose finding period + 42 days maintenance period).

Patients not tolerating their next dose at any time during the 14-days dose finding period will come immediately to the site or call the investigator (unscheduled visit), unless intolerance was detected during a scheduled visit and the dose will be down-titrated to the patient's previous tolerated dose. Then they will continue this treatment for 42 days during the maintenance period.

The dose which will be taken during the maintenance period will be considered as an individual HTD.

I-DM-011SAP 

At the end of the maintenance period, the patient will have the opportunity to continue treatment in an extension study (BIA-51058-202), which is described in a separate protocol.

Patients not tolerating their individual HTD during the maintenance period have to be withdrawn from the study.

#### 2.4 Randomisation

No randomisation will be performed in this study.

#### 2.5 Treatment

The study medication is zamicastat (BIA 5-1058). One tablet of the IMP contains 100 mg of zamicastat.

Each patient will start treatment with 50 mg zamicastat once daily (Dose A) at visit A1 and will be uptitrated step by step to the individual HTD i.e. up to 200 mg zamicastat once daily.

Table 1: Dosage regimen

| Daily dose | |
|------------|------------------------------------------|
| Dose A | 50 mg (half a tablet of 100 mg) |
| Dose B | 100 mg (one tablet of 100 mg) |
| Dose C | 150 mg (one and a half tablet of 100 mg) |
| Dose D | 200 mg (two tablets of 100 mg) |

Each next dose will start after 14 days of treatment if the previous dose was considered safe by the investigator. The up-titration is based on the following safety criteria, including but not limited to:

- Absence of symptomatic and/or clinically relevant orthostatic hypotension
- SBP > 95 mmHg or DBP > 50 mmHg
- Absence of clinically significant changes in ECG parameters (heart rate, P-R interval, QRS duration, QT and QTc interval)
- Absence of clinically significant hypersensitivity/skin allergic reactions

Patients not fulfilling the criteria for up-titration after 14 days of treatment with 50 mg zamicastat have to be withdrawn from the study.

If the patient's next dose will not be tolerated by the patient, the dose has to be down-titrated to his/her previous dose and this dose will be considered as the individual HTD, if tolerated by the patient. Treatment at the individual HTD will be for 42 days during the maintenance period.

Zamicastat has to be taken in the morning after breakfast. The patient must not take the tablet at home on visit days (A3/B3/C3/D3, MPV1, MPV2 and MPV3).

Patients taking 150 mg or 200 mg of zamicastat and who will not participate in the extension study will take 100 mg zamicastat for 14 days.

In case a patient will discontinue the study early due to the occurrence of an AE, down-titration is not mandatory, but at the investigator's discretion.

#### 2.6 Sample Size

The clinical study BIA-51058-201 was designed to explore for the first time the pharmacokinetics, safety and efficacy of zamicastat in PAH patients in its potential therapeutic dose range (50 mg to 200 mg). Since this is an exploratory and descriptive study and no powered comparative statistical analysis is planned, study sample size was not formally calculated. Thus, it was considered that 32 patients constitute an appropriate sample to meet the objectives of the study, considering the low prevalence of the disease and the consequent recruitment constraints.

I-DM-011SAP 

#### Blinding 2.7

Blinding is not applicable to this study.

I-DM-011SAP Effective date: 15.09.2020 

#### 3 ANALYSIS SETS AND SUBGROUPS

#### 3.1 Analysis Sets

Within the framework of this study, the following analysis sets are defined and analysed:

The Enrolled Set (ES) will be defined as all patients who provided informed consent.

The Safety Set (SS) will be defined as all patients who belong to ES with at least one IMP administration.

The Full Analysis Set (FAS) will be defined as all patients who belong to SS with at least one efficacy assessment at visit MPV3.

The modified Full Analysis Set (mFAS) will be defined as all patients who belong to FAS with no substantial changes to their regimen of PAH-approved medications (including diuretics) between visits A1 and MPV3. These patients were defined during Data Review (see Data Review Report, Final 1.0, 10-MAR-2022).

The Pharmacokinetic Analysis Set (PKS) and the Pharmacodynamic (PD) Analysis Set, as well as all corresponding analyses, are described in the reporting and analysis plan prepared by Quotient Sciences Ltd.

Efficacy analyses will be performed on the FAS and mFAS, and the SS will be used for the analysis of the safety endpoints.

#### 3.2 Subgroup Analysis

Subgroups will be formed to explore the effects of right ventricular dysfunction at baseline on selected efficacy parameters based on echocardiography results at V1. The subgroups are described in Table 2 below.

Statistical analyses using subgroups will be conducted when specifically referred to in relevant subsections of Section 5, as not every endpoint might need further evaluation using subgroups.

**Table 2: Subgroup Labels** 

| Number | Description | Label in TLFs |
|--------|-------------------------------------------------|---------------|
| 1 | Right ventricular contractility (TAPSE) ≤ 17 mm | TAPSE ≤ 17 mm |
| 2 | Right ventricular contractility (TAPSE) > 17 mm | TAPSE > 17 mm |

I-DM-011SAP 

## 4 GENERAL DEFINITIONS AND NAMING CONVENTIONS

In order to avoid ambiguity during the analysis, a number of definitions and conventions for data handling are described here.

## 4.1 General Methodology and Presentation of the Results

The default summary statistics for quantitative (continuous) variables will be

- the number of patients (n),
- mean,
- standard deviation (SD),
- coefficient of variation (%CV),
- median.
- minimum (min) and maximum (max)

for patients with data.

Mean and median will be presented to one more decimal place than the raw value. The minimum and maximum values will be presented with the same decimal precision as the raw value. SD will be reported to two decimal places greater than the original value, however no more than 3 decimal places will be presented. CV will be reported to one decimal place.

For qualitative (categorical) variables, the frequency count (n) and percentage (%) of patients with non-missing data per category will be the default frequency tabulations. Where appropriate and present, the number of missing values will be displayed as "Missing" category.

Percentage values are to be presented to one decimal place, for example, 52.3%.

The denominator used for calculation of the percentages will be specified in a footnote to the tables for clarification.

#### 4.2 Statistical Output Layout

All titles and column headers (consisting of one or several words) will be capitalised; articles, prepositions, and conjunctions, and "To" in infinitives will not be capitalised, except they are at the beginning of titles or headers.

All pages will be numbered according to the table/listing/figure to which the page belongs to. Every table/listing/figure will be numbered from page 1, "Page X of Y" at the bottom of each page.

The definition of baseline value will be described in a footnote in every TLF where applicable. Other important definitions will also be presented if necessary.

Dates will be listed in the format: yyyy-mm-dd (e.g. 2003-11-20). Times will be listed in the format: hh:mm (e.g. 09:15) or in the format hh:mm:ss if seconds are collected. When date and time are collected, these are listed in the format: yyyy-mm-ddThh:mm (e.g. 2003-11-20T09:15), yyyy-mm-ddThh, or yyyy-mm-ddThh:mm:ss.

Partial missing dates will be listed in the format yyyy-mm (e.g. 2013-11) if only day is missing or in the format yyyy (e.g. 2013) if month and day are missing.

Missing data including missing dates or times will be displayed in listings as blank fields, unless otherwise specified.

Listings will be sorted by patient's number and visit number where applicable, unless specified otherwise.

## 4.3 Dose Group Names and Labels

Statistical output for baseline characteristics, as well as visit-based safety and efficacy evaluations, will be presented by dose groups. Patients will be allocated to a particular dose group based on their individual HTD, while patients that do not tolerate the 50 mg dose will be allocated to the "No HTD" group for analysis by HTD.

I-DM-011SAP 

Adverse events and concomitant medications will be summarised based on the concurrent IMP dose, without allocating patients to separate dose groups. Details of assignment of concurrent IMP doses will be further described in the Sections 5.3 and 5.6.1.

The labels to be used in the tables, listings and figures are defined in the table below.

**Table 3: Dose Group Labels** 

| Description | Label in TLFs | |
|---|---|---|
| | <b>By Concurrent Dose</b> | By HTD |
| Dose A: 50 mg zamicastat once daily | ZMC 50 mg | No HTD |
| (half a tablet of 100 mg) | | HTD 50 mg |
| Dose B: 100 mg zamicastat once daily | ZMC 100 mg | HTD 100 mg |
| (one tablet of 100 mg) | _ | |
| Dose C: 150 mg zamicastat once daily | ZMC 150 mg | HTD 150 mg |
| (one and a half tablet of 100 mg) | | |
| Dose D: 200 mg zamicastat once daily | ZMC 200 mg | HTD 200 mg |
| (two tablets of 100 mg) | | |

#### 4.4 Visit Names and Labels

This SAP covers only visits which are part of the core study. The extension study (BIA-51058-202) will be covered in a dedicated SAP. The names to be used in the analysis datasets and the labels to be used in the tables, listings and figures for the different study visits are defined below.

**Table 4: Visit Names and Labels** 

| Period Number | | Name | Description | Label in |
|---|---|---|---|---|
| | | | | TLFs |
| Screening | 100 | Visit 1 | Screening visit. Day -12 to -5 | V1 |
| Dose finding | 110 | Visit A1 | Day 1 | A1 |
| | 120 | Visit A2 | 8 days ±2 after A1 (phone call) | A2 |
| | 130 | Visit A3 | 14 days ±2 after A1 | A3 |
| | 220 | Visit B2 | 8 days ±2 after A3 (phone call) | B2 |
| | 230 | Visit B3 | 14 days ±2 after A3 | B3 |
| | 320 | Visit C2 | 8 days ±2 after B3 (phone call) | C2 |
| | 330 | Visit C3 | 14 days ±2 after B3 | C3 |
| | 420 | Visit D2 | 8 days ±2 after C3 (phone call) | D2 |
| | 430 | Visit D3 | 14 days ±2 after C3 | D3 |
| Maintenance 510 Visit MF | | Visit MPV1 | 13 days ±2 after D3/UV for down- | MPV1 |
| | | | titration | |
| | 520 Visit MPV2 | | 27 days ±2 after D3/UV for down- | MPV2 |
| | | | titration | |
| | 530 | Visit MPV3 | 41 days ±2 after D3/UV for down- | MPV3 |
| | | | titration | |
| Dose finding/ 600 Early Discontinua- Wit | | Within 10 days of early | EDV | |
| Maintenance | | tion Visit | discontinuation | |
| Follow-up | | | 14 days ±2 after MPV3/EDV (phone | FUV1 |
| | | [down-titration] call) | | |
| | 620 | Follow-up visit | 14 days ±2 after last IMP intake | FUV2 |

Unscheduled visits (UV) will be numbered and labelled based on the preceding scheduled visit, e.g. "UV A1.1" for the first unscheduled visit after the scheduled visit A1. Multiple unscheduled visits after the same scheduled visit will be numbered and labelled sequentially.

For patients attending the extension study, adverse events and concomitant medications will only be displayed up to the end date of visit MPV3.

I-DM-011SAP 

## 4.5 Day Numbering

All assessment dates will be related to the date of first IMP intake. The date of first IMP intake is referred to as Day 1. Day –1 is the day preceding Day 1 and Day 0 will not be defined. The numbering is such that Day –2 is the day before Day -1, Day 2 is the day after the first IMP intake, etc.

Treatment days may alternatively be numbered with reference to the ongoing study period using the following rules:

- Dates prior to the first IMP intake will be numbered with reference to the date of first IMP intake as described above.
- Dates after the first IMP intake will be numbered with reference to the first day of the ongoing study period using the same rules as described above. Study days during the dose-finding period will be prefixed with the corresponding dose letter (e.g. C-11 for day 11 on the 150 mg dose), study days in the maintenance period will be prefixed with the letter M, and study days in the post-maintenance periods will be prefixed with "DT" and "FU" for the down-titration period and the follow-up period respectively.

For definitions of the study periods, see section 4.6.

## 4.6 Study Periods

### **Screening period**

The Screening period will be defined as the period from informed consent signature date to the first IMP intake date.

#### Dose finding period

The dose finding period will be defined as the period from the date of the first IMP intake to the day before visit D3 or the day before IMP down-titration.

The dose finding period will be split into **dose toleration periods** for each dose prescribed for that period. The period will start from the date of the IMP taken at the site at visit A1/A3/B3/C3 to the day before visit A3/B3/C3/D3 or the day before IMP down-titration.

#### Maintenance period

The maintenance period will be defined as the period between visit D3 or the date of IMP down-titration and the date of the last IMP intake until MPV3 (including the first day of visit). For patients participating in the extension study, the end of the maintenance period will be the end date of visit MPV3.

#### **Down-titration period**

The down-titration period is only applicable to patients not participating in the extension study and with an IMP dispensation at visit MPV3/EDV.

The down-titration period will be defined as the period starting on the second day of MPV3 or one day after visit EDV until the date of the follow-up visit for down titration (FUV1).

## Follow-up period

The follow-up period is only applicable to patients not participating in the extension study.

The follow-up period will be defined as the period between the day after the last IMP intake until the date of study termination.

#### Early discontinuation

For patients who discontinue the study early, the EDV date will be the end date of any ongoing study period.

I-DM-011SAP 

#### 4.7 Baseline Value

#### **Baseline value**

The baseline value for a variable is defined as the last non-missing value collected before the first IMP intake, unless otherwise specified.

See section 5.4.1 Exposure to IMP for definition of first IMP intake.

#### Absolute change from baseline will be calculated as

Absolute Change from Baseline at Visit X = V alue at Visit X - B as line V alue

#### 4.8 Visit Windows

Data will be analysed with the nominal visit number.

## 4.9 Coding Systems and Conventions

## 4.9.1 Coding of adverse events and medical history

Adverse event and medical history investigator terms are assigned to a lowest level term (LLT) and a preferred term (PT) and will be classified by high level term (HLT), high level group term (HLGT) and system organ class (SOC) according to the Medical Dictionary for Regulatory Activities (MedDRA), Version 22.0 or higher.

#### 4.9.2 Coding of medications

Medications are classified according to active drug substance using the WHO Drug Global dictionary, version 2019, March, or higher. The WHO drug code has 11 digits. The generic name is defined by the first 6 of the 11 digits. In addition, the Anatomical Therapeutic Chemical (ATC) classes are assigned to the drug code. In this study, ATC codes are defined to the 4<sup>th</sup> level.

#### 4.10 Handling of Missing Data

No imputations of missing data are planned for this study.

I-DM-011SAP 

# 5 STATISTICAL ANALYSIS: DEFINITIONS, DERIVATIONS, CALCULATIONS AND METHODOLOGY

Protocol no. BIA-51058-201

22-MAR-2022

#### 5.1 Patient Disposition

#### 5.1.1 Disposition and Withdrawals

The following disposition data will be collected in the electronic case report form (eCRF):

- date of informed consent
- date of study termination
- did the patient complete the study as scheduled (yes, no)
- will the patient participate in the extension study (yes, no)
- reason for premature study termination

**Screening failures** will be all patients who have been enrolled in the study (i.e. ICF signed) but discontinue the study before the first IMP intake at visit A1 due to whatever reason (withdrew consent, did not fulfil eligibility criteria, decision of investigator, etc.).

**Withdrawals** will be all patients who have been enrolled and, for whatever reason, discontinue the study after the first IMP intake at visit A1. Patients may withdraw or may be withdrawn from the study for the following reasons:

- At their own request (withdrawal of consent)
- In the investigator's opinion, for reasons of safety or ethics, continuation in the study would be detrimental to the patient's well-being
- Pregnancy
- Ineligibility/development of an exclusion criterion or inclusion criterion no longer fulfilled
- Intolerable adverse event(s)
- At the specific request of the sponsor
- Major protocol deviations
- Patient non-compliance
- Lost to follow up
- Other reasons

Study completion status will be determined by patient's decision to participate in the extension study. If the question "Will the patient participate in the extension study?" in the eCRF is answered as "Yes", the patient will be considered as a completer. If the patient does not participate in the extension study, then the completion status will be based on the Study Termination page in the eCRF.

The following statistical output will be provided:

#### Table 15.1.1.1 Analysis Sets – Enrolled Set

Number and percentage of patients included into the enrolled, safety, full analysis, modified full analysis, pharmacokinetic, and pharmacodynamic analysis sets will be provided.

## Table 15.1.1.2 Reasons for Exclusions from Analysis Sets – Safety Set

Number and percentage of patients excluded from the full analysis, modified full analysis, pharmacokinetic, and pharmacodynamic analysis sets will be provided. Percentages will be based on the number of patients in the safety set. The reasons of exclusion from the analysis sets will be incorporated into the table.

## <u>Table 15.1.2 Screening Failures – Enrolled Set</u>

Counts and percentages of patients who discontinued the study during the screening phase prior to enrolment to the treatment period will be summarised by reasons associated with the discontinuation. Percentage will be based on the number of patients in the enrolled set.

## <u>Table 15.1.4 Patient Disposition – Safety Set</u>

Counts and percentages of patients who completed the treatment period as scheduled, withdrawals during the treatment period will be summarised by HTD and overall. Reasons associated with the termination will be included. Percentage will be based on the number of patients in the safety set.

I-DM-011SAP 

#### Table 15.1.5.1.1 Number of Patients by Country and Site – Enrolled Set

## <u>Table 15.1.5.1.2</u> Number of Patients by Country and Site – Safety Set

Counts and percentages of patients will be presented by country and by site. Percentage will be based on the number of patients in the specified set.

#### Table 15.1.5.2 Number of Patients by Visit – Safety Set

Counts and percentages of patients who continue the study will be presented by visit. Percentage will be based on the number of patients in the safety set.

#### Listing 16.2.1.1.1 Patient Disposition – Safety Set

Patients who enter the treatment period and complete the study as scheduled or as withdrawals will be listed. Reasons for premature study termination will be displayed for withdrawals.

## <u>Listing 16.2.1.1.2 Screening Failures – Enrolled Set</u>

Patients who discontinued the study during the screening phase prior to enrolment to the treatment period will be listed. Reasons associated with the discontinuation will be displayed.

## <u>Listing 16.2.1.2 Patient Visits – Enrolled Set</u>

All visit dates will be listed by patient.

## <u>Listing 16.2.1.4 Exclusions from Analysis Sets – Enrolled Set</u>

Patients excluded from any analysis set and corresponding reasons for exclusion will be listed.

## <u>Figure 15.1.1 Flow Chart of Patient Disposition – Enrolled Set</u>

Number of patients will be displayed in flow chart by their disposition.

## Figure 15.1.2 Flow Chart of Analysis Sets – Enrolled Set

Number of patients will be displayed in flow chart by analysis sets.

#### **5.1.2** Protocol Deviations

Protocol deviations are deviations from the procedures outlined in the clinical study protocol or from subsequent protocol-related instructions like missed evaluations, incorrect timing of evaluations, non-compliance with IMP and intake of prohibited medications or any non-adherence to the clinical study protocol that impacts patient's rights, safety or welfare. Protocol deviations that may affect the pharmacokinetic and pharmacodynamic outcomes will be discussed during the Data Review Meeting (DRM).

In addition, the study disruption due to the COVID-19 pandemic will be assessed in terms protocol deviations and discussed during the DRM. A separate listing for patients affected by the COVID-19 related study disruption will be provided.

Details regarding the DRM will be provided in Section 6.

The following statistical output will be provided:

### Table 15.1.3 Major Protocol Deviations – Safety Set

Number and percentage of patients with major protocol deviations will be summarised by HTD and overall. Protocol deviations will be summarised during the dose finding and maintenance periods and overall. Percentage will be based on the number of patients in the safety set.

## <u>Listing 16.2.1.3.1 Major Protocol Deviations – Safety Set</u>

Patients with major protocol deviations will be listed.

#### Listing 16.2.1.3.2 Patients Affected by the COVID-19 Pandemic – Safety Set

Patients that were affected by the COVID-19 pandemic as well as the details of the deviation will be listed.

#### 5.1.3 Inclusion/Exclusion

The study specific Inclusion/Exclusion Criteria are presented in Section 9.2 and 9.3 of the Clinical Study Protocol.

I-DM-011SAP 

For each criterion, as appropriate, a response of "Yes/No" is to be obtained at Screening and checked again prior to the first IMP administration, at visit A1.

The following statistical output will be provided:

#### Listing 16.2.1.3.3 Inclusion Criteria Not Met and Exclusion Criteria Met - Enrolled Set

Listing of inclusion criteria which were not met and exclusion criteria which were met will be presented per patient.

#### 5.2 Demographic and Other Baseline Characteristics

#### 5.2.1 Demographics

The following demographic characteristics will be presented:

- Age (years)
- Gender (Male, Female)
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Unknown)
- Women of childbearing potential (Yes, No)

Also, the following physical characteristics at baseline will be presented:

- Height (cm)
- Weight (kg)
- Body mass index BMI (kg/m<sup>2</sup>)

Body mass index (BMI) will be calculated as follows:

BMI at Visit X 
$$(kg/m^2) = \frac{Body \ weight \ at \ Visit \ X \ (kg)}{[Body \ height \ at \ Visit \ 1 \ (m)]^2}$$

The following statistical output will be provided:

Table 15.1.6.1.1 Demographics – Safety Set

<u>Table 15.1.6.1.2 Demographics – Full Analysis Set</u>

Table 15.1.6.1.3 Demographics – Pharmacokinetic Analysis Set

Demographic data will be summarised by HTD and overall in the respective set. Percentage for categorical variables will be based on the respective set.

<u>Table 15.1.6.2.1 Baseline Characteristics – Safety Set</u>

Table 15.1.6.2.2 Baseline Characteristics – Full Analysis Set

Table 15.1.6.2.3 Baseline Characteristics – Pharmacokinetic Analysis Set

Weight, height and BMI data will be summarised by HTD and overall in the respective set.

## <u>Listing 16.2.1.5 Demographics and Baseline Characteristics – Enrolled Set</u>

Demographic and baseline characteristic data will be listed for the patients in the enrolled set.

#### **5.2.2** Disease Characteristics

The following information on patient PAH status at baseline will be presented:

- WHO functional class at baseline (see Section 5.5.5)
- The cause of PAH:
  - Idiopathic, in non-vasoreactive patients
  - Heritable: Bone morphogenetic protein receptor type II (BMPR2) mutation and other mutations, in non-vasoreactive patients
  - Drugs and toxin induced, in non-vasoreactive patients
  - Associated with connective tissue disease
  - Associated with simple congenital defects (atrial septal defect and/or ventricular septal defect) if closed > 12 months before inclusion
- Does the patient suffer from scleroderma? (yes, no)

I-DM-011SAP 

The following statistical output will be provided:

Table 15.1.6.3.1 Disease Characteristics – Safety Set

Table 15.1.6.3.2 Disease Characteristics – Full Analysis Set

Table 15.1.6.3.3 Disease Characteristics – Pharmacokinetic Analysis Set

Disease characteristics data will be presented by HTD and overall in the respective set. Percentage for categorical variables will be based on the number of patients in the respective analysis set.

#### <u>Listing 16.2.1.6 Disease Characteristics – Enrolled Set</u>

Disease characteristics data will be listed for the patients in the enrolled set.

## 5.2.3 Medical History

Medical history encompasses relevant prior or ongoing relevant diseases, conditions, hospitalisation and surgical procedures. Medical history records are collected at Visit 1.

Medical history of the patients includes:

- Medical condition/procedure
- Start date
- Stop date
- Ongoing
- Treatment used (yes, no)

Medical history is classified as:

- **Prior medical conditions** are the conditions which started and ended prior to Visit 1.
- **Ongoing medical conditions** are the conditions which are marked as ongoing at Visit 1 or with a stop date at or after Visit 1

In case of partial missing stop dates, a disease will be considered as ongoing at Visit 1, unless the partial date information clearly indicates that the condition stopped prior to Visit 1.

The following statistical output will be provided:

Table 15.1.7.1.1 Prior Medical Conditions - Safety Set

Table 15.1.7.1.2 Prior Medical Conditions - Full Analysis Set

Table 15.1.7.1.3 Prior Medical Conditions - Pharmacokinetic Analysis Set

Table 15.1.7.2.1 Ongoing Medical Conditions – Safety Set

<u>Table 15.1.7.2.2 Ongoing Medical Conditions – Full Analysis Set</u>

Table 15.1.7.2.3 Ongoing Medical Conditions - Pharmacokinetic Analysis Set

Medical history will be summarised displaying counts and percentages of patients having at least one medical condition and will be presented by Primary System Organ Class (SOC) and by Preferred Term (PT) within SOC. SOCs and PT within SOC are to be sorted by descending order of overall incidence. Patients with two or more occurrences of the same condition (as qualified by its PTs) will be counted only once for the respective PT. Percentage will be based on the number of patients in the corresponding analysis set.

## <u>Listing 16.2.1.7 Medical History – Enrolled Set</u>

Medical history conditions will be listed for the patients from the enrolled set

#### 5.3 Prior and Concomitant Medications

Prior and concomitant medications and therapies are documented in the eCRF.

The following information is collected:

- Medication / therapy
- Indication (Medical history condition, Adverse event, Other)
- Total daily dose
- Units

- Route

I-DM-011SAP 

- Frequency
- Start date of medication
- Stop date of medication
- Ongoing (yes, no)

Medications and therapies will be classified as 'prior', 'concomitant' or 'post-treatment' based on start/stop dates:

- **Prior medications/therapies** are defined as those medications/therapies starting and ending prior to the first IMP intake.
- Concomitant medications/therapies are defined as medications/therapies started at or after first IMP intake and include medications/therapies started prior to the first IMP intake but continued during the study.
- **Post-treatment medications/therapies** are defined as medications/therapies which started after the last IMP intake.

If the start or stop date of a medication/therapy is incomplete or missing, it will be assumed to be concomitant except if the incomplete start or stop date indicates that the medication/therapy started and ended prior to the first IMP intake or started after the last IMP intake.

**PAH medications** will be defined as medications where the preferred term for the indication is "pulmonary arterial hypertension", "congenital pulmonary hypertension", or "pulmonary hypertension", as well as any other medications taken for a condition related to PAH. These medications were selected manually during the Data Review (see Data Review Report, Final 1.0, 10-MAR-2022).

In addition, **PAH-approved** medications will be defined as those medications described in the protocol as being an approved PAH therapy (Ambrisentan, Bosentan, Macitentan, Riociguat, Selexipag, Sildenafil, Tadalafil, Epoprostenol intravenous, Iloprost inhaled or Treprostinil intravenous or subcutaneous) and diuretics. PAH-approved medications were selected manually during the Data Review (see Data Review Report, Final 1.0, 10-MAR-2022).

PAH-approved medications will be combined into groups of monotherapy, double therapy, triple therapy, etc., based on the number of PAH-approved medications taken at a given timepoint.

Concomitant medications will be assigned to IMP dose groups based on the prescribed IMP dose at the time of medication intake. If the start or end date indicates that the medication was taken concurrently with multiple doses, it will be assigned to every corresponding dose. If the start or end date is incomplete such that it could belong to more than one dose, the concomitant medication will be assigned to all such doses.

The following statistical output will be provided:

<u>Table 15.1.8.1.1 Prior Medications – Safety Set</u>

Table 15.1.8.1.2 Prior Medications - Full Analysis Set

Table 15.1.8.1.3 Prior Medications – Pharmacokinetic Analysis Set

<u>Table 15.1.8.2.1 Concomitant Medications – Safety Set</u>

Table 15.1.8.2.2 Concomitant Medications – Full Analysis Set

Table 15.1.8.2.3 Concomitant Medications – Pharmacokinetic Analysis Set

The number and percentage of patients with at least one medication within each ATC 2nd level subgroup. Substance name (or combination of substances) will be presented by HTD for prior medication, by dose for concomitant medications and overall in the corresponding analysis set. The ATC 2nd level subgroups and substance drug name within ATC 2nd level subgroup will be ordered by descending overall incidence. Medications that differ at the substance drug name level but belong to the same therapeutic category will be combined.

I-DM-011SAP 

<u>Table 15.1.8.3.1 Prior PAH Medications – Safety Set</u>

Table 15.1.8.3.2 Prior PAH Medications –Full Analysis Set

Table 15.1.8.3.3 Prior PAH Medications – Pharmacokinetic Analysis Set

<u>Table 15.1.8.4.1 Concomitant PAH Medications – Safety Set</u>

<u>Table 15.1.8.4.2 Concomitant PAH Medications – Full Analysis Set</u>

Table 15.1.8.4.3 Concomitant PAH Medications – Pharmacokinetic Analysis Set

Medications for pulmonary arterial hypertension will be summarised as above.

Table 15.1.8.5.1 PAH-Approved Therapy by Visit – Safety Set

Table 15.1.8.5.2 PAH-Approved Therapy by Visit – Full Analysis Set

Table 15.1.8.5.3 PAH-Approved Therapy by Visit – Pharmacokinetic Analysis Set

The number and percentage of patients with PAH-approved monotherapy, double therapy, and triple therapy will be summarised at visits A1 and MPV3. The substance names for each therapy combination will be presented by HTD and overall in the corresponding analysis set.

Listing 16.2.1.8 Medications and Therapies – Enrolled Set

All medications, prior, concomitant and subsequent, will be listed for the patients from the enrolled set.

### 5.4 Exposure to IMP and Compliance

### 5.4.1 Exposure to IMP

Exposure data from the eCRF include:

- First IMP intake
- Last IMP intake before the visit (except unscheduled visits)
- IMP intake at the site (except unscheduled visits)
- Last IMP intake (for withdrawals and patients that do not participate in the extension study)
- Date of IMP down-titration

The overall treatment duration in days will be calculated as follows:

Overall treatment duration (days) = last IMP intake date - first IMP intake date + 1

The following definitions will be used to calculate the overall treatment duration:

- The date of the first IMP intake is the date of the IMP intake as recorded at visit A1.
- The date of the last IMP intake depends on the patient's decision to participate in the extension study. If the patient is not participating in the extension study, then the last IMP intake is the date of the last intake recorded at the study termination page. If the patient is participating in the extension study, then the on-site IMP intake at MPV3 will be the date of the last IMP intake.

The duration of the study periods in days will be calculated as follows:

*Treatment period duration (days)* 

= treatment period end date - treatment period start date + 1

See Section 4.6 for definitions of study periods.

Overall and by-period treatment duration will be adjusted in the case of occurrence of adverse events with associated IMP interruption periods. The calendar days between and including start and stop dates of IMP interruptions will not count towards treatment duration.

The following statistical output will be provided:

<u>Table 15.1.9.1.1 Treatment Duration (days) – Safety Set</u>

Table 15.1.9.1.2 Treatment Duration (days) - Full Analysis Set

<u>Table 15.1.9.1.3 Treatment Duration (days) – Pharmacokinetic Analysis Set</u>

The default summary statistics of treatment duration will be presented by HTD and overall.

I-DM-011SAP 

#### 5.4.2 Compliance

The following compliance-related data will be collected in the eCRF:

- date of IMP dispensation
- prescribed IMP dose
- number of tablets dispensed
- dispensed IMP bottle number
- toleration of IMP dose (Yes, No)
- date of IMP down-titration
- date of IMP return
- number of tablets returned
- returned IMP bottle number

The calculation of the compliance will be based on the total number of tablets prescribed, dispensed and returned overall or during particular study period (for definitions of study periods, see Section 4.6).

22-MAR-2022

The total number of tablets prescribed will be calculated as the prescribed daily number of tablets based on the dose (see Section 2.5) multiplied by the length of the dose prescription in calendar days. The total number of prescribed tablets will be adjusted in the case of occurrence of adverse events with associated IMP interruption periods.

The total number of tablets dispensed and returned will be calculated as the sum of all tablets dispensed and all tablets returned during the corresponding study period. The total number of tablets returned will be considered as missing if not all dispensed bottles are returned in the same corresponding period or the returned bottle(s) is from the previous period.

The overall compliance and compliance during each treatment period will be calculated as:

$$Compliance \ (\%) = \frac{100 \times (tablets \ dispensed - tablets \ returned)}{tablets \ prescribed}$$

In case an IMP bottle is not returned, the overall compliance will be considered as missing.

The following statistical output will be provided:

Table 15.1.9.2.1 Compliance (%) – Safety Set

Table 15.1.9.2.2 Compliance (%) - Full Analysis Set

Table 15.1.9.2.3 Compliance (%) – Pharmacokinetic Analysis Set

The default summary statistics of compliance will be presented by HTD and overall for the respective analysis set. Number and percentage of patients will also be summarised by compliance categories  $(< 90\%, \ge 90\% \text{ and } \le 110\%, \ge 110\%)$  for the respective analysis set.

## <u>Listing 16.2.2.1 Drug Accountability – Safety Set</u>

Information related drug accountability will be listed for the patients from the safety set.

#### <u>Listing 16.2.2.2 Exposure to IMP and Compliance – Safety Set</u>

Information related exposure to IMP and compliance will be listed for the patients from the safety set.

I-DM-011SAP 

#### 5.5 Analysis of Efficacy Endpoints

The following efficacy related secondary endpoints will be calculated and analysed:

- Right heart catheterisation parameters
- 6-MWT, including Borg dyspnoea score
- Biomarker (NT-proBNT)
- Echocardiogram parameters
- NYHA/WHO functional class
- Quality of life (SF-36v2)

Efficacy data will be analysed exploratively. Continuous measures will be summarised using summary statistics, in addition for the changes from baseline a 95% confidence interval will be provided. Categorical variables will be summarised by using frequency counts and percentages.

## 5.5.1 Right Heart Catheterisation

Right heart catheterisation (RHC) will be performed at visit A1 and at visit MPV3 before IMP intake to determine the change of haemodynamic parameters in the patients. If available, results from a right heart catheterisation within 90 days before V1 may be used in place of the V1 measurement. The following haemodynamic parameters will be collected:

- Cardiac output (L/min) (CO)
- Mixed venous oxygen saturation (%)  $(S_vO_2)$
- Pulmonary artery pressure systolic (mmHg) (PAPs)
- Pulmonary artery pressure diastolic (mmHg) (PAPd)
- Mean pulmonary artery pressure (mmHg) (mPAP)
- Pulmonary artery wedge pressure (mmHg) (PAWP)
- Right atrial pressure (mmHg) (RAP)
- Transpulmonary pressure gradient (mmHg) (**TPG**)
- Diastolic pressure gradient (mmHg) (**DPG**)
- Pulmonary vascular resistance (dyn\*s/cm<sup>5</sup>) (PVR)
- Systemic ventricular resistance (dyn\*s/cm<sup>5</sup>) (SVR)
- Cardiac index (L/min/m<sup>2</sup>) (CI)
- Pulmonary arterial compliance (mL/mmHg) (PAC, SV/PP)
- Heart rate (bpm)
- Stroke volume (mL/beat) (SV)
- Stroke volume index (mL/m²/beat) (SVI)

The derived parameters mPAP, TPG, DPG, PVR, PAC, SV, and SVI will be recalculated from other parameters using standardised formulae below.

$$mPAP = PAPd + (PAPs - PAPd)/3$$
  
 $TPG = mPAP - PAWP$   
 $DPG = PAPd - PAWP$   
 $PVR = (mPAP - PAWP)/CO \cdot 80$   
 $PAC = SV/(PAPs - PAPd)$   
 $SV = CO/HR \cdot 1000$   
 $SVI = CI/HR \cdot 1000$ 

The recalculated parameter values will be used in summaries and listings.

The clinical significance (yes/no) of any abnormal right heart catheterisation findings will be assessed by the investigator.

**Post-DR note:** Clinical significance as assessed by the investigator will not be used for statistical analyses (see Data Review Report, Final 1.0, 10-MAR-2022). Instead, right heart catheterisation results

I-DM-011SAP 

will be assigned a "Low", "Normal" or "High" value according to ranges defined by Table 4. The ranges are based on the Data Validation Plan (Final 3.0, 21-JUL-2020).

**Table 5: Right Heart Catheterisation Normal Ranges** 

| Parameter | Normal Range |
|---|---|
| Cardiac output (L/min) (CO) | 2.5-8.0 |
| Mixed venous oxygen saturation (%) (S <sub>v</sub> O <sub>2</sub> ) | 60-80 |
| Pulmonary artery pressure systolic (mmHg) (PAPs) | 25-80 |
| Pulmonary artery pressure diastolic (mmHg) (PAPd) | 8-16 |
| Mean pulmonary artery pressure (mmHg) (mPAP) | ≥25 |
| Pulmonary artery wedge pressure (mmHg) (PAWP) | ≤15 |
| Right atrial pressure (mmHg) (RAP) | <14 |
| Transpulmonary pressure gradient (mmHg) (TPG) | >12 |
| Diastolic pressure gradient (mmHg) (DPG) | >6 |
| Pulmonary vascular resistance (dyn*s/cm <sup>5</sup> ) (PVR) | 250-1000 |
| Systemic vascular resistance (dyn*s/cm <sup>5</sup> ) (SVR) | 800-1200 |
| Cardiac index (L/min/m²) (CI) | >2 |
| Pulmonary arterial compliance (mL/mmHg) (PAC; SV/PP) | 0.4-3.8 |
| Heart rate (bpm) | 50-100 |
| Stroke volume (mL/beat) (SV) | >50 |
| Stroke volume index (mL/m²/beat) (SVI) | >30 |

Recalculated results will be used for applicable parameters.

The following statistical output will be provided:

<u>Table 15.2.1.1.4 Summary of Right Heart Catheterization Parameters – Modified Full Analysis Set</u>
The default summary statistics of RHC test results will be presented by HTD and overall at visits A1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

# <u>Table 15.2.1.1.5 Summary of Right Heart Catheterization Parameters – Modified Full Analysis Set</u> (TAPSE Subgroups)

The default summary statistics of RHC parameters PVR, mPAP, RAP, and CI will be presented by TAPSE subgroup and overall at visits A1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

<u>Table 15.2.1.2.1 Incidence of Right Heart Catheterisation Abnormalities – Full Analysis Set Table 15.2.1.2.2 Incidence of Right Heart Catheterisation Abnormalities – Modified Full Analysis Set Number and percentage of patients with abnormal values will be displayed by HTD and overall in not CS abnormal and CS abnormal categories. Percentage will be based on the number of patients at specified visit.</u>

<u>Table 15.2.1.3.1 Shift Table of Right Heart Catheterisation Results – Full Analysis Set Table 15.2.1.3.2 Shift Table of Right Heart Catheterisation Results – Modified Full Analysis Set Shift tables showing changes in the number and frequency of patients in not CS abnormal and CS abnormal categories between baseline and MPV3 will be provided.</u>

<u>Listing 16.2.3.1 Right Heart Catheterisation Parameters – Enrolled Set</u> Values of parameters of right heart catheterisation will be listed.

I-DM-011SAP 

### 5.5.2 6-Min Walk Test (6-MWT)

The 6-MWT is a self-paced test of walking capacity used to assess aerobic capacity and endurance. It plays a key role in evaluation functional exercise capacity, assessing prognosis and evaluating response to treatment across a wide range of respiratory diseases. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

The test will be performed at visit V1 before IMP intake and at visit MPV3 before right heart catheterisation.

At screening, two attempts must be performed, separated by at least 30 minutes. The attempt in which the longer distance was covered will be considered as baseline. In case the distance covered during both attempts is equal, the first attempt will be considered as baseline.

The following parameters will be collected:

- SpO<sub>2</sub> (%) before and after the test
- Borg Dyspnoea score before and after the test
- Heart rate (bpm) before and after the test
- Lap length (m)
- Number of laps completed
- Distance covered (m)
- Time walking (min)
- Oxygen flow rate (L/min)
- Number of stops
- Time stopped (min)

The Borg Dyspnoea score is a patient-reported measure for assessing breathlessness. Symptoms of breathlessness are rated on a scale of 0-10, where 0 indicates no symptoms and 10 indicates the most severe breathlessness.

The differences in SpO<sub>2</sub>, the Borg Dyspnoea score, and heart rate between after and before the test will be calculated. These differences will be displayed as additional parameters in summaries.

The following statistical output will be provided:

Table 15.2.2.1 Summary of 6-MWT by HTD – Full Analysis Set

Table 15.2.2.2 Summary of 6-MWT – Full Analysis Set

Table 15.2.2.3 Summary of 6-MWT by HTD – Modified Full Analysis Set

Table 15.2.2.4 Summary of 6-MWT - Modified Full Analysis Set

The default summary statistics of 6-MWT test results will be presented by HTD and overall at visits V1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

#### Table 15.2.2.5 Summary of 6-MWT Distance – Modified Full Analysis Set (TAPSE Subgroups)

The default summary statistics of 6-MWT distance travelled will be summarised by TAPSE subgroup and overall at visits V1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

## <u>Listing 16.2.3.2-Min Walk Test – Enrolled Set</u>

Values of parameters of 6-Min walk test will be listed.

I-DM-011SAP 

#### 5.5.3 Biomarker

Blood samples will be collected for biomarker NT-proBNP (pg/mL) evaluation at visits V1 and MPV3. NT-proBNP will be summarized in the unit ng/L for statistical output. No derivations are needed as the conversion factor between these units is 1.

The following statistical output will be provided:

Table 15.2.3.1.1 Summary of Biomarker NT-proBNP (ng/L) by HTD – Full Analysis Set

Table 15.2.3.1.2 Summary of Biomarker NT-proBNP (ng/L) – Full Analysis Set

Table 15.2.3.1.3 Summary of Biomarker NT-proBNP (ng/L) by HTD – Modified Full Analysis Set

Table 15.2.3.1.4 Summary of Biomarker NT-proBNP (ng/L) – Modified Full Analysis Set

The default summary statistics of biomarker NT-proBNP will be presented by HTD and overall at visits V1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

<u>Table 15.2.3.2.1 Summary of Biomarker NT-proBNP (ng/L) by Pooled HTD –Full Analysis Set</u>
<u>Table 15.2.3.2.2 Summary of Biomarker NT-proBNP (ng/L) by Pooled HTD – Modified Full Analysis Set</u>
<u>Set</u>

Biomarker NT-proBNP will be summarised as above, with HTD pooled into "HTD < 200 mg" and "HTD 200 mg" groups.

<u>Figure 15.2.1.1 Box-Whisker Plot of NT-proBNP by Pooled HTD – Full Analysis Set Figure 15.2.1.2 Box-Whisker Plot of NT-proBNP by Pooled HTD – Modified Full Analysis Set Box-whisker plots of NT-proBNP will be displayed by HTD at visits V1 and MPV3. The HTD will be pooled into "HTD < 200 mg" and "HTD 200 mg" groups. Summary statistics will be displayed below each box.</u>

<u>Listing 16.2.3.3 Biomarker NT-proBNP – Enrolled Set</u>

Values of biomarker NT-proBNP will be listed.

#### 5.5.4 Echocardiography

Transthoracic echocardiography is used to image the effects of PAH on the heart. An echocardiogram (ECHO) will be performed at Visit 1 and MPV3.

The following parameters will be determined:

- Tricuspid regurgitation (absent, mild, moderate or severe)
- Right ventricular contractility (TAPSE) (mm)
- Pericardial effusion (absent, traces or present)
- Right atrial area (end-systolic) (cm<sup>2</sup>)
- Right ventricular end-diastolic area (cm<sup>2</sup>)

The clinical significance (yes/no) of any abnormal ECHO findings will be assessed by the investigator.

The following statistical output will be provided:

<u>Table 15.2.4.1.1 Summary of Categorical Echocardiography Parameters – Full Analysis Set</u>
<u>Table 15.2.4.1.2 Summary of Categorical Echocardiography Parameters – Modified Full Analysis Set</u>
Number and percentage of patients will be displayed by HTD and overall at visits V1 and MPV3.

Percentage will be based on the number of patients at the specified visit.

<u>Table 15.2.4.2.4 Summary of Numerical Echocardiography Parameters – Modified Full Analysis Set</u> The default summary statistics of ECHO parameters will be presented by HTD and overall at visits V1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

I-DM-011SAP 

# Statistical Analysis Plan, Version Final 1.0

## Table 15.2.4.2.5 Summary of Numerical Echocardiography Parameters – Modified Full Analysis Set (TAPSE Subgroups)

The default summary statistics of ECHO parameters will be presented by TAPSE subgroup and overall at visits V1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

## Table 15.2.4.3.1 Incidence of Echocardiography Abnormalities – Full Analysis Set

### Table 15.2.4.3.2 Incidence of Echocardiography Abnormalities – Modified Full Analysis Set

Number and percentage of patients will be displayed by HTD and overall in Not CS abnormal and CS abnormal categories. Percentage will be based on the number of patients at the specified visit.

### Table 15.2.4.4.1 Shift Table of Echocardiography Results – Full Analysis Set

## Table 15.2.4.4.2 Shift Table of Echocardiography Results – Modified Full Analysis Set

Shift tables showing changes in the number and frequency of patients in Not CS abnormal and CS abnormal categories between V1 and MPV3 visits will be provided.

#### Listing 16.2.3.4 Echocardiography – Enrolled Set

Values of echocardiography tests will be listed.

#### New York Heart Association/Word Health Organisation Functional Class 5.5.5 (NYHA/WHO)

Classification of functional status of patients will be performed at Visit 1 and at visit MPV3/EDV by the investigator by using the NYHA/WHO classification system defined below.

#### **Table 6:NYHA/WHO Classes**

| Class | Description |
|---|---|
| Class I | Patients with pulmonary hypertension but without resulting limitation of physical |
| | activity. Ordinary physical activity does not cause undue dyspnoea or fatigue, chest |
| | pain or near syncope. |
| Class II | Patients with pulmonary hypertension resulting in a slight limitation of physical |
| | activity. They are comfortable at rest. Ordinary physical activity causes undue |
| | dyspnoea or fatigue, chest pain or near syncope. |
| Class III | Patients with pulmonary hypertension resulting in marked limitation of physical |
| | activity. They are comfortable at rest. Less than ordinary activity causes undue |
| | dyspnoea or fatigue, chest pain or near syncope. |
| Class IV | Patients with pulmonary hypertension with inability to carry out any physical activity |
| | without symptoms. These patients' manifest signs of right heart failure. Dyspnoea |
| | and/or fatigue may even |

The following statistical output will be provided:

## Table 15.2.5.1.1 Summary of NYHA/WHO Functional Class – Full Analysis Set

## Table 15.2.5.1.2 Summary of NYHA/WHO Functional Class – Modified Full Analysis Set

Number and percentage of patients will be displayed by HTD and overall in each NYHA/WHO functional class. Percentage will be based on the number of patients at the specified visit.

## Table 15.2.5.2.1 Shift Table of NYHA/WHO Functional Class – Full Analysis Set

## Table 15.2.5.2.2 Shift Table of NYHA/WHO Functional Class – Modified Full Analysis Set

Shift tables showing changes in the number and frequency of patients with respect to the NYHA/WHO functional class between V1 and MPV3/EDV will be provided.

#### Listing 16.2.3.5 NYHA/WHO Functional Class – Enrolled Set

NYHA/WHO functional class data will be listed by visit.

#### Quality of Life (SF-36v2) 5.5.6

The 36-item Short Form Survey version 2 (SF-36v2) is used to assess the quality of life. The questionnaire will be completed by the patient at Visit 1 and at MPV3.

I-DM-011SAP 

SF-36v2 asks 36 questions (items) to measure functional health and well-being from the patient's point of view. All but one (question 2) of the 36 items will be used to score the eight SF-36v2 health domains:

- Physical Functioning (PF)
- Role Limitations due to Physical Health (RP)
- Bodily Pain (BP)
- General Health (GH)
- Vitality (VT)
- Social Functioning (SF)
- Role Limitations due to Emotional Health (RE)
- Mental Health (MH).

A total score will be calculated for each SF-36v2 health domain by taking the sum of the corresponding responses and rescaling it to a range of 0 to 100, where 100 represents the best possible result. Each domain will then be standardised using a general population norm.

The scores of the eight health domains will be used to calculate a physical component summary (PCS) and mental component summary (MCS) score using coefficients based on a principal components analysis of the SF-36v2 domain scores in the general population. The PCS and MCS are summary measures that represent the overall physical and mental health of the patient, with higher scores representing better outcomes.

A subset of items from six domains (PF, RE, SF, BP, MH, VT) will be used to calculate a Utility Index Score, which rates the overall health state from 0.0 (worst health state) to 1.0 (best health state). The updated (SF-6D R2) Utility Index Score will be summarised.

Optum PRO CoRE will be used to generate the following scores:

- SF-36v2 domain scores (0-100 scale)
- SF-36v2 domain scores based on the 2009 US general population norms
- PCS and MCS scores based on the 2009 US general population norms
- SF-6D R2

In addition, interpretations for the norm-based SF-36v2 health domains and PCS and MCS scores will be provided based on benchmarks from the general population cardiac patients:

- "Well Below", if the norm-based score is 10 points or more below the benchmark;
- "Below", if the norm-based score is from 5 to 9 points below the benchmark;
- "Same or Better", if the norm-based score is less than 5 points below the benchmark.

The following statistical output will be provided:

Table 15.2.6.1.1 Summary of SF-36v2 Domain Scores by HTD – Full Analysis Set

Table 15.2.6.1.2 Summary of SF-36v2 Domain Scores – Full Analysis Set

Table 15.2.6.1.3 Summary of SF-36v2 Domain Scores by HTD – Modified Full Analysis Set

Table 15.2.6.1.4 Summary of SF-36v2 Domain Scores – Modified Full Analysis Set

The default summary statistics of SF-36v2 results will be presented by HTD and overall at visits V1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

<u>Table 15.2.6.2.1 Summary of Norm-Based SF-36v2 Domain Scores by HTD – Full Analysis Set</u>

Table 15.2.6.2.2 Summary of Norm-Based SF-36v2 Domain Scores-Full Analysis Set

Table 15.2.6.2.3 Summary of Norm-Based SF-36v2 Domain Scores by HTD – Modified Full Analysis Set

Table 15.2.6.2.4 Summary of Norm-Based SF-36v2 Domain Scores – Modified Full Analysis Set
The default summary statistics of SF-36v2 results based on 2009 US norms will be presented by HTD and overall at visits V1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

I-DM-011SAP 

Table 15.2.6.3.1 Summary of SF-36v2 Utility Index Scores by HTD – Full Analysis Set

Table 15.2.6.3.2 Summary of SF-36v2 Utility Index Scores – Full Analysis Set

Table 15.2.6.3.3 Summary of SF-36v2 Utility Index Scores by HTD - Modified Full Analysis Set

Table 15.2.6.3.4 Summary of SF-36v2 Utility Index Scores – Modified Full Analysis Set

The default summary statistics of Utility Index scores will be presented by HTD and overall at visits V1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

Table 15.2.6.4.1 Summary of SF-36v2 Cardio Benchmark Interpretation – Full Analysis Set

<u>Table 15.2.6.4.2 Summary of SF-36v2 Cardio Benchmark Interpretation – Modified Full Analysis Set</u> Number and percentage of patients will be displayed by HTD at visits V1 and MPV3. Percentage will be based on the number of patients at the specified visit.

<u>Table 15.2.6.5.1 Shift Table of SF-36v2 Cardio Benchmark Interpretation – Full Analysis Set</u>
<u>Table 15.2.6.5.2 Shift Table of SF-36v2 Cardio Benchmark Interpretation – Modified Full Analysis Set</u>
Shift tables showing changes in the number and frequency of patients with respect to the Cardio benchmark interpretation between V1 and MPV3 will be provided.

Figure 15.2.2.1 Norm-Based SF-36v2 Domain Scores by Visit – Full Analysis Set

Figure 15.2.2.2 Norm-Based SF-36v2 Domain Scores by Visit – Modified Full Analysis Set

The means of norm-based SF-36v2 domain scores will be presented by HTD at visits V1 and MPV3 using a bar chart. A reference line will be included for the average score in the general population.

Figure 15.2.3.1 SF-36v2 Cardio Benchmark Interpretation by Visit – Full Analysis Set

<u>Figure 15.2.3.2 SF-36v2 Cardio Benchmark Interpretation by Visit – Modified Full Analysis Set</u>

The numbers of patients in each cardio benchmark interpretation category will be displayed by HTD for each domain at visits V1 and MPV3 using a stacked bar chart.

<u>Listing 16.2.3.6 SF-36v2 – Enrolled Set</u>

Summary scores based on the SF-36v2 survey results will be listed.

#### 5.6 Analysis of Safety Endpoints

Safety will be assessed by evaluation of the following variables:

- Adverse events
- Clinically relevant changes in laboratory parameters (haematology, biochemistry, coagulation, urinalysis, arterial blood gas analysis)
- Clinically relevant changes in vital signs
- Clinically relevant changes in ECG
- Physical examination findings
- Number of digital scars (only in patients with scleroderma)
- Modified Rodnan Skin score (only in patients with scleroderma)

#### **5.6.1** Adverse Events

AEs will be coded according to latest Medical Dictionary for Regulatory Activities (MedDRA®) Version 22.0.

Adverse events' data include:

- adverse event name
- start/stop dates
- ongoing
- severity (mild, moderate, severe)
- relationship (not related, unlikely, possible, probable, definite)
- action taken with study medication (dose not changed, dose reduced, drug interrupted, drug withdrawn, not applicable, unknown)
- other actions (none, medication required, tests required, withdrawn from the study, hospitalisation required or prolonged, other specification)

I-DM-011SAP 

- Protocol no. BIA-51058-201 22-MAR-2022
- outcome of event (recovered/resolved, recovering/resolving, not recovered/not resolved, recovered/resolved with sequelae, fatal, unknown)
- AE of special interest (yes or no)
- seriousness (yes or no)
- start/stop dates of drug interruption

All AEs will be presented in listings.

Summaries of adverse events will include AEs defined as **treatment-emergent adverse events** (**TEAEs**), defined as AEs with the first onset or worsening after the first IMP intake and not more than 14 days after the last IMP intake.

If the start date of an AE is incomplete or missing, it will be assumed to be treatment-emergent except if the incomplete start date or the stop date indicates that the event started or ended prior to the first IMP intake or started later than 14 days after last IMP intake.

AEs will be further assigned to the following categories:

- Serious Adverse Events (SAEs): defined as AEs considered by the investigator as serious.
- Adverse Event of Special Interest (AESIs): defined as AEs assessed by the investigator as being of special interest.
- **Related TEAEs**: defined as AEs assessed as being "Possible", "Probable" or "Definite" to IMP and include the events with missing IMP relationship assessment.
- **Unrelated TEAEs**: defined as AEs assessed as being "Not related" or "Unlikely" to be related to IMP.
- **Severe TEAEs**: defined as AEs assessed as being "Severe" in intensity and include the events with missing severity assessment.
- **TEAEs leading to down-titration:** defined as AEs where "Action taken with study medication" is indicated as "dose reduced".
- **TEAEs leading to discontinuation:** selected as those events where "Action taken with study medication" is indicated as "drug withdrawn" or "other actions" is "discontinued from study".
- **TEAEs leading to death:** selected as those events where outcome of event is indicated as "fatal".

Adverse events will be assigned to IMP dose groups based on the prescribed IMP dose at the date of AE onset. AEs with an onset date on the same day as a down-titration will be assigned to the previous dose. If the AE onset date is incomplete such that it could belong to more than one prescribed dose, the AE will be assigned to all such doses.

The following statistical output will be provided:

#### Table 15.3.1.1 Overall Summary of TEAEs – Safety Set

An overview of TEAEs:

- TEAE
- Non-serious TEAE
- Serious TEAE
- TEAEs of special interest
- Related TEAE
- Related serious TEAE
- Mild TEAE
- Moderate TEAE
- Severe TEAE
- TEAE leading to down-titration
- TEAE leading to discontinuation
- Serious TEAE leading to discontinuation

I-DM-011SAP 
- Related TEAE leading to discontinuation
- TEAE leading to death

will be displayed during the trial as well as the dose finding, maintenance, and down-titration periods by dose and overall for the patients in the safety set.

Table 15.3.1.2 Incidence of TEAEs – Safety Set

Table 15.3.1.3 Incidence of Serious TEAEs – Safety Set

Table 15.3.1.4 Incidence of TEAEs of Special Interest – Safety Set

Table 15.3.1.5 Incidence of Related TEAEs - Safety Set

<u>Table 15.3.1.6 Incidence of Related Serious TEAEs – Safety Set</u>

Table 15.3.1.7 Incidence of TEAEs Leading to Down-Titration – Safety Set

<u>Table 15.3.1.8 Incidence of TEAEs Leading to Discontinuation – Safety Set</u>

Table 15.3.1.9 Incidence of TEAEs Leading to Death – Safety Set

TEAEs occurring during the trial as well as the dose finding, maintenance, and down-titration periods will be summarised by concurrent dose and overall via the numbers of adverse events, as well as counts and percentages of patients having experienced adverse events during the dose finding and maintenance periods and overall. Percentages will be based on the number of patients in the safety set. Here and in the tables below the SOCs and PTs within each SOC will be ordered by descending overall incidence.

In addition, the following will be provided summarised by SOC and PT for the safety set for each dose and overall:

Table 15.3.1.10 Incidence of TEAEs by Severity – Safety Set

Table 15.3.1.11 Incidence of TEAEs by Relationship to IMP – Safety Set

All adverse event data will be listed as follows:

Listing 16.2.4.1.1 Adverse Events: MedDRA Coding

Listing 16.2.4.1.2 Adverse Events: General – Enrolled Set

Listing 16.2.4.1.3 Non-Serious Adverse Events – Safety Set

Listing 16.2.4.1.4 Serious Adverse Events – Safety Set

Listing 16.2.4.1.5 TEAEs of Special Interest – Safety Set

<u>Listing 16.2.4.1.6 AEs Leading to Discontinuation – Safety Set</u>

<u>Listing 16.2.4.1.7 AEs Leading to Death – Safety Set</u>

All AEs will be displayed by patient including the PT of an AE, start and stop dates, duration and other characteristics of AEs.

#### **5.6.2** Clinical Laboratory Evaluation

Clinical laboratory values for haematology, coagulation, biochemistry and urinalysis will be collected at screening (V1), visits A3/B3/C3/D3, MPV1, MPV3/EDV and FUV2 for each laboratory parameter.

Blood pregnancy test values will be collected only for women with childbearing potential at screening (V1) and urine pregnancy test will be collected at visits A1, A3/B3/C3/D3, MPV1, MPV2, MPV3/EDV and FUV2. For patients enrolled under protocol version final 1.0, urine pregnancy test will be evaluated at visits A1, A3/B3/C3/D3, MPV1, MPV2, MPV3/EDV.

The following parameters will be collected:

- Haematology: haemoglobin, haematocrit, red blood cell count (RBC), white blood cell count (WBC), differential - neutrophils, eosinophils, lymphocytes, monocytes and basophils, and platelet count.
- Coagulation: prothrombin time test (INR).
- **Biochemistry:** sodium, potassium, chloride, calcium, phosphate, blood urea nitrogen, aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), lactate dehydrogenase (LDH), alkaline phosphatase (ALP), creatine phosphokinase (CPK), creatinine, glucose, C-reactive protein, albumin, total protein, total cholesterol, low-density lipoprotein-cholesterol, high-density lipoprotein-cholesterol, triglycerides, and total bilirubin (bilirubin will be fractionated direct/indirect if elevated), haemoglobin A1c (HbA1c).

I-DM-011SAP 

Statistical Analysis Plan, Version Final 1.0

Urinalysis: pH, specific gravity, protein, blood, glucose, ketones, bilirubin, urobilinogen, leucocytes and nitrites (local dipstick). Microscopy and other appropriate tests (as needed) will be performed if dipstick indicates any relevant abnormality.

Haematology, coagulation and biochemistry test results will be assigned an LNH classification according to whether the value is lower than (L), within (N) or higher than (H) the reference range for that parameter as provided by the corresponding laboratory.

For urinalysis shift tables, all parameters except pH and specific gravity will be assigned a "normal"/"abnormal" category based on the recorded result. "Negative" and "normal" results will be considered as normal, and any positive results will be considered as abnormal.

Clinical significance of laboratory values will be evaluated by the investigator.

The following statistical output will be provided:

Table 15.3.2.1.1.1 Summary of Clinical Laboratory Tests: Haematology by HTD- Safety Set

Table 15.3.2.1.1.2 Summary of Clinical Laboratory Tests: Haematology – Safety Set

Table 15.3.2.1.2.1 Summary of Clinical Laboratory Tests: Biochemistry by HTD – Safety Set

Table 15.3.2.1.2.2 Summary of Clinical Laboratory Tests: Biochemistry – Safety Set

Table 15.3.2.1.3.1 Summary of Clinical Laboratory Tests: Coagulation by HTD – Safety Set

Table 15.3.2.1.3.2 Summary of Clinical Laboratory Tests: Coagulation – Safety Set

The default summary statistics of clinical laboratory test results will be presented by HTD and overall at V1, A3/B3/C3/D3, MPV1, MPV3/EDV and FUV2. The absolute change from baseline will be presented as well.

Table 15.3.2.1.4 Summary of Clinical Laboratory Tests: Urinalysis – Safety Set

Number and percentage of patients will be displayed by HTD and overall at V1, A3/B3/C3/D3, MPV1, MPV3/EDV and FUV2. Percentage will be based on the number of patients at the specified visit.

Table 15.3.2.2.1 Clinical Laboratory Tests: Incidence of Haematology Abnormalities – Safety Set

Table 15.3.2.2.2 Clinical Laboratory Tests: Incidence of Biochemistry Abnormalities – Safety Set

Table 15.3.2.2.3 Clinical Laboratory Tests: Incidence of Coagulation Abnormalities – Safety Set

Number and percentage of patients for each laboratory parameter will be displayed by HTD and overall in Low, CS Low, Normal, High and CS High categories. Percentage will be based on the number of patients at specified visit.

Table 15.3.2.2.4 Clinical Laboratory Tests: Incidence of Urinalysis Abnormalities – Safety Set

Number and percentage of patients for each laboratory parameter will be displayed by HTD and overall in Normal, Abnormal and CS abnormal categories. Percentage will be based on the number of patients at specified visit.

Table 15.3.2.3.1 Clinical Laboratory Tests: Shift Table of Haematology Results – Safety Set

Table 15.3.2.3.2 Clinical Laboratory Tests: Shift Table of Biochemistry Results - Safety Set

Table 15.3.2.3.3 Clinical Laboratory Tests: Shift Table of Coagulation Results – Safety Set

Shift tables showing changes in the number and frequency of patients with respect to the normal range between baseline and MPV3/EDV will be provided.

Table 15.3.2.3.4 Clinical Laboratory Tests: Shift Table of Urinalysis Results – Safety Set

Shift tables showing changes in the number and frequency of patients in Normal, Abnormal and CS abnormal categories between baseline and MPV3/EDV will be provided.

Listing 16.2.4.2.1 Laboratory Data: Haematology – Enrolled Set

Listing 16.2.4.2.2 Laboratory Data: Biochemistry – Enrolled Set

<u>Listing 16.2.4.2.3 Laboratory Data: Coagulation – Enrolled Set</u>

Values of laboratory tests will be listed.

<u>Listing 16.2.4.2.4 Laboratory Data: Urinalysis – Enrolled Set</u>

All urinalysis (dipstick) data will be listed.

Listing 16.2.4.2.5 Laboratory Data: Microscopy – Enrolled Set

All microscopy data will be listed.

I-DM-011SAP 

#### Protocol no. BIA-51058-201 22-MAR-2022

# <u>Listing 16.2.4.2.6 Laboratory Data: Pregnancy Tests – Enrolled Set</u>

Data of pregnancy tests will be listed.

#### 5.6.3 Arterial Blood Gas Analysis

Arterial blood gas analysis will be performed at visit A1 and MPV3 before first IMP intake.

The following parameters of Arterial blood gas analysis will be collected:

- Fraction of inspired oxygen (%) (FiO<sub>2</sub>)
- pH
- oxygen partial pressure (mmHg) (pO<sub>2</sub>)
- carbon dioxide partial pressure (mmHg) (pCO<sub>2</sub>)
- bicarbonate (mEq/L)
- base excess (mEq/L) (BE)
- arterial oxygen saturation (%) (SaO<sub>2</sub>)\*
- sodium (mEq/L)
- potassium (mEq/L)
- lactate (mEq/L)
- \* Collected as "O2 content (%)" in earlier eCRF versions.

If arterial blood gas analysis is not performed, then peripheral oxygen saturation (%) will be collected.

The clinical significance (yes/no) of any abnormal Arterial blood gas analysis findings will be assessed by the investigator. Parameter values without a clinical significance evaluation will be considered as "Normal", and values with "No" or "Yes" clinical significance evaluations will be considered as "NCS Abnormal" and "CS Abnormal", respectively.

The following statistical output will be provided:

#### Table 15.3.3.1.1 Summary of Arterial Blood Gas Analysis by HTD – Safety Set

## Table 15.3.3.1.2 Summary of Arterial Blood Gas Analysis – Safety Set

The default summary statistics of Arterial blood gas analysis parameters will be presented by HTD and overall at visits A1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

# <u>Table 15.3.3.2 Incidence of Arterial Blood Gas Analysis Abnormalities – Safety Set</u>

Number and percentage of patients with abnormal values will be displayed by HTD and overall in Not CS abnormal and CS abnormal categories. Percentage will be based on the number of patients at specified visit.

# Table 15.3.3.3 Shift Table of Arterial Blood Gas Analysis Results – Safety Set

Shift tables showing changes in the number and frequency of patients in Not CS abnormal and CS abnormal categories between baseline and MPV3/EDV will be provided.

# Table 15.3.3.4.1 Summary of Peripheral Oxygen Saturation (%) by HTD – Safety Set

# Table 15.3.3.4.2 Summary of Peripheral Oxygen Saturation (%) – Safety Set

The default summary statistics of peripheral oxygen saturation (%) will be presented by HTD and overall at visits A1 and MPV3. The absolute change from baseline will be presented as well. For the changes from baseline a 95% confidence interval will be provided.

### <u>Listing 16.2.4.3 Arterial blood gas analysis – Enrolled Set</u>

Values of arterial blood gas analysis and peripheral oxygen saturation (%) will be listed.

## 5.6.4 Vital Signs

Vital signs will be collected at screening (V1), visits A1, A3/B3/C3/D3, MPV1, MPV2, MPV3/EDV and FUV2. Blood pressure and heart rate will be measured in supine position (two measurements) and afterwards in standing position (one measurement). Tympanic body temperature will also be assessed.

I-DM-011SAP 

At visits A1 and MPV3, blood pressure and heart rate will be measured before IMP intake as well as 4, 8 and 24 hours after IMP intake. For patients enrolled under protocol version final 1.0, vital signs were only evaluated before IMP intake.

Systolic and diastolic blood pressure and pulse rate will be summarised by measurement position. The mean value of measurements in the supine position at a given timepoint will be used in summaries. **Orthostatic changes** in vital sign parameters will also be calculated as the difference between the measurement in the standing position and the mean of the supine measurements. The orthostatic changes will be displayed after each corresponding parameter's standing position results in summaries.

To evaluate the short-term effects of the IMP on vital sign parameters, the absolute change from the pre-dose value within the corresponding visit will be calculated for each parameter at visits A1 and MPV3. Additionally, the difference in the within-visit changes will be evaluated for each corresponding timepoint between visits MPV3 and A1.

**Physical measurements** – height and weight will be assessed at visit V1. Weight will also be measured at MPV3/EDV. BMI will be calculated from available data (see Section 5.2.1 for calculation).

The following statistical output will be provided:

## Table 15.3.4.1.1 Summary of Vital Signs by HTD- Safety Set

#### Table 15.3.4.1.2 Summary of Vital Signs – Safety Set

Vital sign parameters will be summarised including change from baseline at each timepoint by HTD and overall.

## <u>Table 15.3.4.2 Summary of Vital Signs by Pooled HTD – Safety Set</u>

Vital sign parameters will be summarised as above, with HTD pooled into "HTD < 200 mg" and "HTD 200 mg" groups.

# Table 15.3.4.3.1 Summary of Short-Term IMP Effect on Vital Signs by HTD – Safety Set

## Table 15.3.4.3.2 Summary of Short-Term IMP Effect on Vital Signs – Safety Set

The observed values and absolute changes from the pre-dose value will be summarised for each vital sign parameter at each timepoint by HTD and overall.

# <u>Table 15.3.4.4.1 Summary of Change in Short-Term IMP Effect on Vital Signs by HTD – Safety Set</u> Table 15.3.4.4.2 Summary of Change in Short-Term IMP Effect on Vital Signs – Safety Set

The changes from pre-dose values and the differences in changes from pre-dose values will be summarised between corresponding timepoints at visits A1 and MPV3 by HTD and overall.

# Table 15.3.4.5.1 Summary of Physical Measurements by HTD – Safety Set

#### Table 15.3.4.5.2 Summary of Physical Measurements – Safety Set

Physical measurements will be summarised including change from baseline at each timepoint by HTD and overall.

#### Figure 15.3.1 Vital Signs Median Change from Baseline – Safety Set

The median changes from baseline of vital signs parameters at each post-baseline timepoint will be displayed by will be displayed by HTD. The HTD will be pooled into "HTD < 200 mg" and "HTD 200 mg" groups.

#### Listing 16.2.4.4 Vital Signs and Physical Measurements – Enrolled Set

Values of vital signs and physical measurements will be listed.

# 5.6.5 12-Lead Electrocardiogram (ECG) Data

A simultaneous 12-lead resting electrocardiogram (ECG) will be collected at screening (V1), A1, A3/B3/C3/D3, MPV1, MPV2, MPV3/EDV and FUV2. At visits A1 and MPV3 triplicate ECG recordings will be performed at following time points - before IMP intake as well as 4 and 8 hours after IMP intake. At EDV only one ECG recording will be performed. For patients enrolled under protocol version final 1.0, ECG assessments were only collected once at visits V1, A3/B3/C3/D3, MPV1, MPV3/EDV.

Following parameters will be assessed:

I-DM-011SAP 

- Heart rate (bpm)
- P-R interval (msec)
- ORS duration (msec)
- QTcF interval (msec)
- QT interval (msec)
- P pulmonale
- Right axis deviation
- RV hypertrophy
- RV strain
- Right bundle branch block
- Heart rhythm (normal, abnormal)

For patients enrolled under protocol version final 1.0, heart rhythm was not collected.

Clinical significance (yes/no) of any abnormal ECG data findings will be assessed by the investigator. Parameter values without a clinical significance evaluation will be considered as "Normal", and values with "No" or "Yes" clinical significance evaluations will be considered as "NCS Abnormal" and "CS Abnormal", respectively.

Where multiple ECG recordings are performed within a visit or timepoint, ECG parameters will be summarised as follows. For numeric parameters, the mean of collected values will be used in summaries. For abnormality assessments, the worst value within the visit/timepoint will be used.

To evaluate the short-term effects of the IMP on ECG parameters, the absolute change from the predose value within the corresponding visit will be calculated for each parameter at visits A1 and MPV3. Additionally, the difference in the within-visit changes will be evaluated for each corresponding timepoint between visits MPV3 and A1.

The following statistical output will be provided:

#### Table 15.3.5.1.1 Summary of ECG Assessments by HTD – Safety Set

## <u>Table 15.3.5.1.2 Summary of ECG Assessments – Safety Set</u>

ECG parameters will be summarised including change from baseline at each visit by HTD and overall.

# <u>Table 15.3.5.2.1 Summary of Short-Term IMP Effect on ECG Assessments by HTD – Safety Set</u>

#### Table 15.3.5.2.2 Summary of Short-Term IMP Effect on ECG Assessments – Safety Set

The observed values and absolute changes from the pre-dose value will be summarised for each vital sign parameter at each timepoint by HTD and overall.

# <u>Table 15.3.5.3.1 Summary of Change in Short-Term IMP Effect on ECG Assessements by HTD – Safety Set</u>

<u>Table 15.3.5.3.2 Summary of Change in Short-Term IMP Effect on ECG Assessements – Safety Set</u>
The changes from pre-dose values and the differences in changes from pre-dose values will be summarised between corresponding timepoints at visits A1 and MPV3 by HTD and overall.

# Table 15.3.5.4.1 Incidence of ECG Abnormalities – Safety Set

Number and percentage of patients with Not CS abnormal and CS abnormal ECG parameters assessments will be displayed by HTD and overall. Percentage will be based on the number of patients at specified visit.

#### Table 15.3.5.4.2 Shift Table of ECG Abnormalities – Safety Set

Shift tables showing changes in the number and frequency of patients in not CS abnormal and CS abnormal categories between baseline and MPV3/EDV will be provided. The worst abnormality assessment collected during MPV3/EDV will be selected for each patient. Percentage will be based on the number of patients in the safety set.

#### Table 15.3.5.4.3 Shift Table of Within-Visit ECG Abnormalities – Safety Set

Shift tables showing changes in the number and frequency of patients in not CS abnormal and CS abnormal categories between the pre-dose measurement and each post-dose measurement at each visit.

I-DM-011SAP 

Protocol no. BIA-51058-201 22-MAR-2022

The worst abnormality assessment collected during the corresponding timepoint will be selected for each patient. Percentage will be based on the number of patients in the safety set.

## <u>Listing 16.2.4.5 Electrocardiogram – Enrolled Set</u>

Values of simultaneous 12-lead resting electrocardiogram tests will be listed.

## 5.6.6 Physical Examination Findings

Physical examinations will be performed at Visit 1, visits A3/B3/C3/D3, MPV1, MPV2, MPV3/EDV on relevant body systems (appearance, skin, eyes, ears-nose-throat, lungs-chest, heart, abdomen, extremities, other). Clinical significance (yes/no) of any abnormal physical examination findings and specification of clinically significant abnormality findings will be assessed by the investigator.

The following statistical output will be provided:

#### <u>Table 15.3.6 Summary of Physical Examination Findings – Safety Set</u>

Number and percentage of patients with not CS abnormal and CS abnormal physical examinations findings will be displayed at each visit by HTD and overall. Percentage will be based on the number of patients at the specified visit.

#### Listing 16.2.4.6 Physical Examinations – Enrolled Set

Values of physical examination will be listed.

#### 5.6.7 Number of Digital Scars

Number of digital scars will be documented in patients with scleroderma only.

At Visit 1 the investigator will document the number of existing digital scars at the fingers and toes. At visits A3/B3/C3/D3, MPV1, MPV2 and MPV3/EDV the investigator will examine fingers and toes of the patient and will document the number of digital scars. Additionally, the clinical examination will be supported by interviewing the patient.

For patients enrolled with protocol version 1.0 the investigator documented only the number of new scars at post-baseline visits, therefore the total number of scars will be derived adding number of scars at baseline and new scars.

The following statistical output will be provided:

# <u>Table 15.3.7.1 Summary of Scleroderma Scarring by HTD – Safety Set</u>

#### Table 15.3.7.2 Summary of Scleroderma Scarring – Safety Set

The default summary statistics of number of digital scars will be presented by HTD and overall at each visit. The absolute change from baseline will be presented as well.

# <u>Listing 16.2.4.7 Number of Digital Scars – Enrolled Set</u>

Number of scars will be listed by visit.

#### 5.6.8 Modified Rodnan Skin Score (mRSS)

The mRSS is a measure of skin thickness and is used as an outcome measure for scleroderma.

The score consists of an evaluation of patient's skin thickness rated by clinical palpation using a scale from 0 to 3 (0=normal skin; 1=mild thickness; 2=moderate thickness; 3=severe thickness) for each of 17 surface anatomic areas of the body: face, anterior chest, abdomen, (right and left separately) fingers, forearms, upper arms, tights, lower legs, dorsum of hands and feet. These individual values are added, and the sum is defined as the total skin score.

The investigator will document the total skin score at Visit 1 and visit MPV3/EDV.

I-DM-011SAP 

**Protocol no. BIA-51058-201** 22-MAR-2022

The following statistical output will be provided:

Table 15.3.8.1 Summary of mRSS by HTD – Safety Set

<u>Table 15.3.8.2 Summary of mRSS – Safety Set</u>

The default summary statistics of modified Rodnan score will be presented by HTD and overall at each visit. The absolute change from baseline will be presented as well.

<u>Listing 16.2.4.8 Modified Rodnan Skin Score – Enrolled Set</u>

Values of mRSS will be listed.

I-DM-011SAP 

# 6 DATA REVIEW

The aims of the Data Review (DR) are:

- to identify major/minor protocol deviations, that may affect the pharmacokinetic or pharmacodynamic outcomes, or the treatment of the patients
- to identify impacts of the COVID-19 pandemic on the study conduct
- to solve any outstanding issues in the SAP
- to discuss any open data issues

The DR will be performed after data entry and following a database lock. All decisions made during the DR will be documented in the DR report before the closure of the database.

An appropriate clinical study team, including a physician, will review potential protocol deviations and relevant information regarding those deviations to determine a possible impact on pharmacokinetic endpoints. The status, major or minor, of each protocol deviation will be documented in the DR report. A patient may have one or more major protocol deviations resulting in the exclusion of that patient from the PKS set.

Protocol deviations will, if possible, be validated against data recorded in the eCRF. Where an answer for an inclusion/exclusion tick box differs from the algorithmic check of the criteria, the algorithmic check will overrule the tick box.

Additionally, protocol deviations will be reviewed by the medical monitor and will be categorized according to their impact on the PK analysis into following groups: major, minor and case by case decision.

Protocol deviations of the following categories and respective data listings will be reviewed during the DR.

# **Inclusion Criteria**

| No. | Inclusion Criteria Deviation | Major/ |
|---|---|---|
| | | Minor/ |
| | | Case by |
| | | case review |
| PD#01. | Male or female patients aged 18 to 75 years, inclusive. | Case by case |

Protocol Versions Final 1.0 and 2.0:

Male or female patients aged 18 to 65 years.

PD#02. Able to comprehend and willing to sign an informed consent form (ICF). Major

PD#03. Diagnosis of PAH (pulmonary arterial hypertension WHO Group 1) Case by case documented by RHC with a mPAP ≥ 25 mmHg, a PAWP ≤ 15 mmHg and a PVR > 3 WU [8,9]:

- a) Idiopathic, in non-vasoreactive patients
- b) Heritable: Bone morphogenetic protein receptor type II (BMPR2) mutation and other mutations, in non-vasoreactive patients
- c) Drugs and toxin induced, in non-vasoreactive patients
- d) Associated with connective tissue disease
- e) Associated with simple congenital defects (atrial septal defect and/or ventricular septal defect) if closed > 12 months before inclusion.

PD#04. Added in Protocol Version Final 3.0:

Minor

Protocol no. BIA-51058-201

22-MAR-2022

The patient's last right heart catheterisation results, which were measured at the study site, must not be older than 90 days before V1 (will be considered as baseline value). Otherwise a right heart catheterisation has to be performed as part of the study at visit A1.

I-DM-011SAP 

Protocol no. BIA-51058-201 22-MAR-2022

#### **No.** Inclusion Criteria Deviation

Major/ Minor/ Case by case review

PD#05. WHO functional class II or III as judged by the investigator.

Case by case

PD#06. Stable treatment with at least one of the following approved PAH therapies for at least 90 days prior to V1: Ambrisentan, Bosentan, Macitentan, Riociguat, Selexipag, Sildenafil, Tadalafil, Epoprostenol intravenous, Iloprost inhaled or Treprostinil intravenous or subcutaneous.

Case by case

Protocol Version Final 1.0:

Stable treatment with at least one of the following approved oral PAH therapies within 3 months before V1: Ambrisentan, Bosentan, Macitentan, Riociguat, Selexipag, Sildenafil or Tadalafil.

PD#07. Added in Protocol Version Final 3.0:

Minor

For women: Agree not to donate ova from the time of informed consent until 30 days after the last IMP intake.

For men: Agree not to donate sperm from the time of informed consent until 90 days after the last IMP intake.

#### **Exclusion Criteria**

# No. Exclusion Criteria Deviation

Major/ Minor/ Case by case review

PD#08. Contraindication to zamicastat, i.e. known hypersensitivity to ingredients of zamicastat formulation.

Minor

PD#09. Two or more consecutive measurements of SBP < 95 mmHg or DBP < 50 M mmHg measured at V1.

Minor

Protocol Version Final 2.0

Two or more consecutive measurements of SBP  $\leq$  95 mmHg or DBP  $\leq$  50 mmHg.

Protocol Version Final 1.0:

Persistent hypotension defined as SBP < 95 mmHg or DBP < 50 mmHg.

PD#10. Uncontrolled diabetes mellitus with HbA1c ≥ 8.5% within the last three Minor months or at screening.

Protocol Version Final 1.0:

Uncontrolled diabetes mellitus.

PD#11. PAH WHO Group 1 due to portal hypertension, human immunodeficiency Case by case virus (HIV) infection and schistosomiasis.

PD#12. Any disease known to cause pulmonary hypertension other than PAH WHO Case by case Group 1.

Protocol Version Final 1.0:

Any disease known to cause pulmonary hypertension other than PAH WHO Group 1 e.g. obstructive lung diseases, parasitic disease affecting the pulmonary system, sickle cell anaemia, left heart disease.

PD#13. Added in Protocol Version Final 2.0:

Case by case


#### Protocol no. BIA-51058-201

#### **No.** Exclusion Criteria Deviation

Major/ Minor/ Case by case review

22-MAR-2022

Obstructive lung disease: Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC) < 60% and FEV1 < 60% of predicted value after bronchodilator administration.

PD#14. Restrictive lung disease: Total Lung Capacity (TLC) < 70% of predicted value, as demonstrated and documented by previous spirometry data which, in the opinion of the investigator, represent the clinical state of the patient at the time of the screening visit.

Case by case

Added in Protocol Version Final 2.0:

Restrictive lung disease: Total Lung Capacity (TLC) < 70% of predicted value.

- PD#15. History of moderate to severe hepatic impairment (Child-Pugh B and C). Case by case
- PD#16. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m<sup>2</sup> Case by case (measured at V1).
- PD#17. Use of the following prohibited medication or treatments during study participation: calcium channel blockers (CCBs) if used for the treatment of PAH in vasoreactive patients; drugs containing a catechol group that is metabolised by DβH e.g. rimiterole, isoprenaline, dopamine, dopexamine or dobutamide or α- and/or β-blockers.
- PD#18. Current or previous (within the past year) alcohol or substance abuse Minor excluding caffeine or nicotine.

Case by case

PD#19. Presence of any other significant or progressive/unstable medical condition that, in the opinion of the investigator, would compromise evaluation of the study treatment or may jeopardise the patient's safety, compliance or adherence to protocol requirements.

Minor

PD#20. For women: Pregnancy or breast-feeding. Women of childbearing potential (as defined in Section 4.2) unable or unwilling to undergo pregnancy tests and practice highly effective contraceptive measures in combination with a barrier method condom (without spermicidal foam/gel/film/cream/suppository or fat- or oil-containing lubricants), occlusive cap (diaphragm or cervical/vault caps) with spermicidal gel/film/cream/suppository from the time of informed consent until 30 days after last IMP intake. Highly effective methods for women are surgical intervention (e.g. bilateral tubal occlusion), non-hormonal implantable intrauterine device, true sexual abstinence (i.e. when this is in line with the preferred and usual lifestyle of the patient) and vasectomised partner (provided that the partner is the sole sexual partner of the patient and the partner has received medical assessment of the surgical success). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods), hormonal contraceptives and withdrawal are not acceptable methods of contraception.

For men: Male patients who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved acceptable contraceptive measure from the time of informed consent until 90 days after the last IMP intake. The following methods are acceptable methods of contraception: partner's use of combined (oestrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); partner's use of progestogen-only hormonal contraception (oral, injectable/implantable,

I-DM-011SAP 

# No. Exclusion Criteria Deviation

Major/ Minor/ Case by case review

22-MAR-2022

Protocol no. BIA-51058-201

intrauterine hormone-releasing system); partner's use of implantable intrauterine device; surgical sterilisation (for example, vasectomy or bilateral tubal occlusion).

#### Protocol Version Final 2.0:

For women: Pregnancy or breast-feeding. Women of childbearing potential unable or unwilling to undergo pregnancy tests and practice acceptable contraceptive measures from the time of informed consent until 30 days after last IMP intake. Acceptable methods for women are surgical intervention (e.g. bilateral tubal occlusion), non-hormonal implantable intrauterine device, double-barrier methods, true sexual abstinence (i.e. when this is in line with the preferred and usual lifestyle of the patient) and vasectomised partner (provided that the partner is the sole sexual partner of the patient and the partner has received medical assessment of the surgical success). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), hormonal contraceptives and withdrawal are not acceptable methods of contraception.

For men: Male patients who are sexually active with a partner of childbearing potential must use, with their partner, a condom plus an approved acceptable contraceptive measure from the time of informed consent until 90 days after the last IMP intake. The following methods are acceptable methods of contraception: partner's use of combined (oestrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); partner's use of progestogen-only hormonal contraception (oral, injectable/implantable, intrauterine hormone-releasing system); partner's use of implantable intrauterine device; surgical sterilisation (for example, vasectomy or bilateral tubal occlusion).

#### Protocol Version Final 1.0:

For women: Pregnancy or breast-feeding. Women of childbearing potential unable or unwilling to undergo pregnancy tests and practice acceptable contraceptive measures. Acceptable methods for women are surgical intervention (e.g. bilateral tubal occlusion), intrauterine device, double-barrier methods and true sexual abstinence (i.e. when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

PD#21. Previous participation in any other drug investigational study within the C past 30 days (or five half-lives of investigational medicinal product [IMP] whichever is longer) prior to V1.

Case by case

PD#22. Vulnerable patients according to Section 1.61 of the ICH guideline for Minor Good Clinical Practice E6

I-DM-011SAP 

# **Additional Study Conduct Deviations**

| No. | Deviation | Major/<br>Minor/<br>Case by |
|---|---|---|
| PD#23. | Down-titration dose not according to the protocol. | case review<br>Case by<br>case |
| PD#24. | Up-titration safety criteria deviations | Minor |
| PD#25. | IMP compliance <90% or >110% by period or overall | Case by case |
| PD#26. | Schedule deviations of visits with scheduled IMP dispensations | Case by case |
| PD#27. | Time deviations of scheduled assessments (ECG, Vital signs, blood withdrawal for PK/PD) at A1 and MPV3 | Case by case |
| PD#28. | Deviations in sequences of assessments/tests/procedures | Minor |
| PD#29. | Prohibited medications/therapies | Case by case |
| PD#30. | Adverse events with possible impact on primary endpoint. | Case by case |
| PD#31. | Missing/incomplete blood withdrawal for PK, blood and urinalysis sampling for PD | Case by case |
| PD#32. | Missing/incomplete test/examination assessments: | Minor |
| | vital signs, physical measurements, NYHA/WHO functional class, laboratory tests, physical examination, ECG, number of digital scars, modified Rodnan Skin Score, SF-36v2, 6-min walk test, echocardiography, right heart catheterisation, blood withdrawal biomarker | |
| PD#33. | Protocol deviations documented by CRAs and selected by medical monitors for discussion during DR | Case by case |

Protocol no. BIA-51058-201

22-MAR-2022

Reference listings will be made available to help with the review of the protocol deviations. The specific content and format of listings to be reviewed during the DR meeting (including any additional requirements that may be necessary to aid in review) will be determined outside the scope of this SAP.

#### 7 INTERIM ANALYSIS

No interim analysis is planned for this study.

I-DM-011SAP 

# **Protocol no. BIA-51058-201** 22-MAR-2022

# 8 CHANGES TO THE ANALYSIS AS LAID DOWN IN THE PROTOCOL AND AMENDMENTS

No changes to the analysis as laid down in the clinical study protocol and protocol amendment(s) were made.

I-DM-011SAP 

#### 9 REFERENCES

- 1. SAS® Institute Inc., Cary, North Carolina, United States of America, Version 9.4.
- 2. MedDRA Medical Dictionary for Regulated Activities. International Federation of Pharmaceutical Manufacturers Associations (IFPMA), c/o TRW, VAR1/8A/MSSO, 12011 Sunset Hills Road, Reston, VA 20190-3285, USA, Version 22.0, 1 March 2019.
- 3. WHODrug Global dictionary. World Health Organization Collaborating Center for International Drug Monitoring, P.O. Box 26, S-751 03 Uppsala, Sweden, version 2019, March
- 4. Optum, Inc 1301 Atwood Avenue, Suite 311 N Johnston, R.I. 02919, U.S.A, Pro Core Version 1.4

I-DM-011SAP 

#### 10 APPENDICES

The following documents are attached as appendices to the SAP:

- 1. 0223\_TableShells\_1.0\_20220322.docx
- 2. 0223\_ListingShells\_1.0\_20220322.docx
- 3. 0223 FigureShells 1.0 20220322.docx
- 4. QSC202579 (BIA-51058-201) RAP\_20Feb2020\_Finalv1.0.pdf

# 10.1 Tables

Appendix tables defined below will be provided in separate .rtf files for each output.

| No | Table Identifier, Title | Output file |
|---|---|---|
| Dem | Demographic and Study Population Data | |
| 1 | Table 15.1.1.1 Analysis Sets – Enrolled Set | BIA-T-150101010000-anlset-enr.rtf |
| 2 | Table 15.1.1.2 Reasons for Exclusion from Analysis<br>Sets – Safety Set | BIA-T-150101020000-reas-excl-ss.rtf |
| 3 | Table 15.1.2 Screening Failures – Enrolled Set | BIA-T-150102000000-scrfail-enr.rtf |
| 4 | Table 15.1.3 Major Protocol Deviations – Safety Set | BIA-T-150103000000-protdev-ss.rtf |
| 5 | Table 15.1.4 Patient Disposition – Safety Set | BIA-T-150104000000-disp-ss.rtf |
| 6 | Table 15.1.5.1.1 Number of Patients by Country and Site – Enrolled Set | BIA-T-150105010100-countrysite-enr.rtf |
| 7 | Table 15.1.5.1.2 Number of Patients by Country and Site – Safety Set | BIA-T-150105010200-countrysite-ss.rtf |
| 8 | Table 15.1.5.2 Number of Patients by Visit – Safety Set | BIA-T-150105020000-visits-ss.rtf |
| 9 | Table 15.1.6.1.1 Demographics – Safety Set | BIA-T-150106010100-dm-ss.rtf |
| 10 | Table 15.1.6.1.2 Demographics – Full Analysis Set | BIA-T-150106010200-dm-fas.rtf |
| 11 | Table 15.1.6.1.3 Demographics – Pharmacokinetic Analysis Set | BIA-T-150106010300-dm-pks.rtf |
| 12 | Table 15.1.6.2.1 Baseline Characteristics – Safety Set | BIA-T-150106020100-basechar-ss.rtf |
| 13 | Table 15.1.6.2.2 Baseline Physical Characteristics – Full Analysis Set | BIA-T-150106020200-basechar-fas.rtf |
| 14 | Table 15.1.6.2.3 Baseline Physical Characteristics – Pharmacokinetic Analysis Set | BIA-T-150106020300-basechar-pks.rtf |
| 15 | Table 15.1.6.3.1 Disease Characteristics – Safety Set | BIA-T-150106030100-diseasechar-ss.rtf |
| 16 | Table 15.1.6.3.2 Disease Characteristics – Full Analysis Set | BIA-T-150106030200-diseasechar-fas.rtf |
| 17 | Table 15.1.6.3.3 Disease Characteristics – Pharmacokinetic Analysis Set | BIA-T-150106030300-diseasechar-pks.rtf |
| 18 | Table 15.1.7.1.1 Prior Medical Conditions – Safety Set | BIA-T-150107010100-mh-prior-ss.rtf |
| 19 | Table 15.1.7.1.2 Prior Medical Conditions – Full Analysis Set | BIA-T-150107010200-mh-prior-fas.rtf |
| 20 | Table 15.1.7.1.3 Prior Medical Conditions –<br>Pharmacokinetic Analysis Set | BIA-T-150107010300-mh-prior-pks.rtf |
| 21 | Table 15.1.7.2.1 Ongoing Medical Conditions – Safety Set | BIA-T-150107020100-mh-ongoing-ss.rtf |
| 22 | Table 15.1.7.2.2 Ongoing Medical Conditions – Full Analysis Set | BIA-T-150107020200-mh-ongoing-fas.rtf |
| 23 | Table 15.1.7.2.3 Ongoing Medical Conditions –<br>Pharmacokinetic Analysis Set | BIA-T-150107020300-mh-ongoing-pks.rtf |
| 24 | Table 15.1.8.1.1 Prior Medications – Safety Set | BIA-T-150108010100-priormed-ss.rtf |
| 25 | Table 15.1.8.1.2 Prior Medications – Full Analysis Set | BIA-T-150108010200-priormed-fas.rtf |
| 26 | Table 15.1.8.1.3 Prior Medications – Pharmacokinetic Analysis Set | BIA-T-150108010300-priormed-pks.rtf |
| 27 | Table 15.1.8.2.1 Concomitant Medications – Safety Set | BIA-T-150108020100-conmed-ss.rtf |

I-DM-011SAP 

| 28 | Table 15.1.8.2.2 Concomitant Medications – Full Analysis Set | BIA-T-150108020200-conmed-fas.rtf |
|---|---|---|
| 29 | Table 15.1.8.2.3 Concomitant Medications – Pharmacokinetic Analysis Set | BIA-T-150108020300-conmed-pks.rtf |
| 30 | Table 15.1.8.3.1 Prior PAH Medications – Safety Set | BIA-T-150108030100-priormed-pah-ss.rtf |
| 31 | Table 15.1.8.3.2 Prior PAH Medications – Full Analysis Set | BIA-T-150108030200-priormed-pah-fas.rtf |
| 32 | Table 15.1.8.3.3 Prior PAH Medications – Pharmacokinetic Analysis Set | BIA-T-150108030300-priormed-pah-pks.rtf |
| 33 | Table 15.1.8.4.1 Concomitant PAH Medications – Safety Set | BIA-T-150108040100-conmed-pah-ss.rtf |
| 34 | Table 15.1.8.4.2 Concomitant PAH Medications – Full Analysis Set | BIA-T-150108040200-conmed-pah-fas.rtf |
| 35 | Table 15.1.8.4.3 Concomitant PAH Medications – Pharmacokinetic Analysis Set | BIA-T-150108040300-conmed-pah-pks.rtf |
| 36 | Table 15.1.8.5.1 PAH-Approved Therapy by Visit – Safety Set | BIA-T-150108050100-pahappr-byvis-ss.rtf |
| 37 | Table 15.1.8.5.2 PAH-Approved Therapy by Visit – Full Analysis Set | BIA-T-150108050200-pahappr-byvis-fas.rtf |
| 38 | Table 15.1.8.5.3 PAH-Approved Therapy by Visit – Pharmacokinetic Analysis Set | BIA-T-150108050300-pahappr-byvis-<br>pks.rtf |
| 39 | Table 15.1.9.1.1 Treatment Duration (days) – Safety Set | BIA-T-150109010100-trtdur-ss.rtf |
| 40 | Table 15.1.9.1.2 Treatment Duration (days) – Full Analysis Set | BIA-T-150109010200-trtdur-fas.rtf |
| 41 | Table 15.1.9.1.3 Treatment Duration (days) –<br>Pharmacokinetic Analysis Set | BIA-T-150109010300-trtdur-pks.rtf |
| 42 | Table 15.1.9.2.1 Compliance (%) – Safety Set | BIA-T-150109020100-compl-ss.rtf |
| 43 | Table 15.1.9.2.2 Compliance (%) – Full Analysis Set | BIA-T-150109020200-compl-fas.rtf |
| 44 | Table 15.1.9.2.3 Compliance (%) – Pharmacokinetic Analysis Set | BIA-T-150109020300-compl-pks.rtf |
| Effic | eacy Data | |
| 45 | Table 15.2.1.1.1 Summary of Right Heart Catheterisation Parameters by HTD – Full Analysis Set | BIA-T-150201010100-rhc-htd-fas.rtf |
| 46 | Table 15.2.1.1.2 Summary of Right Heart<br>Catheterization Parameters – Full Analysis Set | BIA-T-150201010200-rhc-tot-fas.rtf |
| 47 | Table 15.2.1.1.3 Summary of Right Heart Catheterisation Parameters by HTD – Modified Full Analysis Set | BIA-T-150201010300-rhc-htd-mfas.rtf |
| 48 | Table 15.2.1.1.4 Summary of Right Heart Catheterization Parameters – Modified Full Analysis Set | BIA-T-150201010400-rhc-tot-mfas.rtf |
| 49 | Table 15.2.1.1.5 Summary of Right Heart Catheterization Parameters – Modified Full Analysis Set (TAPSE Subgroups) | BIA-T-150201010500-rhc-tapse-mfas.rtf |
| 50 | Table 15.2.1.2.1 Incidence of Right Heart Catheterisation Abnormalities – Full Analysis Set | BIA-T-150201020100-rhc-abnorm-fas.rtf |
| 51 | Table 15.2.1.2.2 Incidence of Right Heart Catheterisation Abnormalities – Modified Full Analysis Set | BIA-T-150201020200-rhc-abnorm-mfas.rtf |
| 52 | Table 15.2.1.3.1 Shift Table of Right Heart Catheterisation Results – Full Analysis Set | BIA-T-150201030100-rhc-shift-fas.rtf |
| 53 | Table 15.2.1.3.2 Shift Table of Right Heart Catheterisation Results – Modified Full Analysis Set | BIA-T-150201030200-rhc-shift-mfas.rtf |
| 54 | Table 15.2.2.1 Summary of 6-MWT by HTD – Full Analysis Set | BIA-T-150202010000-6mwt-htd-fas.rtf |
| | | t |
| 55 | Table 15.2.2.2 Summary of 6-MWT – Full Analysis<br>Set | BIA-T-150202020000-6mwt-tot-fas.rtf |
| 56 | Set Table 15.2.2.3 Summary of 6-MWT by HTD – | BIA-T-150202020000-6mwt-tot-fas.rtf BIA-T-150202030000-6mwt-htd-mfas.rtf |
| | Set | |

I-DM-011SAP 

| 58 | Table 15.2.2.5 Summary of 6-MWT Distance – Modified Full Analysis Set (TAPSE Subgroups) | BIA-T-150202050000-6mwt-tapse-mfas.rtf |
|---|---|---|
| 59 | Table 15.2.3.1.1 Summary of Biomarker NT-proBNP (ng/L) by HTD – Full Analysis Set | BIA-T-150203010100-biomarker-htd-fas.rtf |
| 60 | Table 15.2.3.1.2 Summary of Biomarker NT-proBNP (ng/L) – Full Analysis Set | BIA-T-150203010200-biomarker-tot-fas.rtf |
| 61 | Table 15.2.3.1.3 Summary of Biomarker NT-proBNP (ng/L) by HTD – Modified Full Analysis Set | BIA-T-150203010300-biomarker-htd-<br>mfas.rtf |
| 62 | Table 15.2.3.1.4 Summary of Biomarker NT-proBNP (ng/L) – Modified Full Analysis Set | BIA-T-150203010400-biomarker-tot-<br>mfas.rtf |
| 63 | Table 15.2.3.2.1 Summary of Biomarker NT-proBNP (ng/L) by Pooled HTD –Full Analysis Set | BIA-T-150203020100-biomarker-htdpool-<br>fas.rtf |
| 64 | Table 15.2.3.2.2 Summary of Biomarker NT-proBNP (ng/L) by Pooled HTD – Modified Full Analysis Set | BIA-T-150203020200-biomarker-htdpool-<br>mfas.rtf |
| 65 | Table 15.2.4.1.1 Summary of Categorical<br>Echocardiography Parameters– Full Analysis Set | BIA-T-150204010100-echo-cat-fas.rtf |
| 66 | Table 15.2.4.1.2 Summary of Categorical Echocardiography Parameters – Modified Full Analysis Set | BIA-T-150204010200-echo-cat-mfas.rtf |
| 67 | Table 15.2.4.2.1 Summary of Numerical<br>Echocardiography Parameters by HTD – Full Analysis<br>Set | BIA-T-150204020100-echo-num-htd-fas.rtf |
| 68 | Table 15.2.4.2.2 Summary of Numerical<br>Echocardiography Parameters – Full Analysis Set | BIA-T-150204020200-echo-num-tot-fas.rtf |
| 69 | Table 15.2.4.2.3 Summary of Numerical Echocardiography Parameters by HTD – Modified Full Analysis Set | BIA-T-150204020300-echo-num-htd-mfas.rtf |
| 70 | Table 15.2.4.2.4 Summary of Numerical<br>Echocardiography Parameters – Modified Full<br>Analysis Set | BIA-T-150204020400-echo-num-tot-mfas.rtf |
| 71 | Table 15.2.4.2.5 Summary of Numerical<br>Echocardiography Parameters – Modified Full<br>Analysis Set (TAPSE Subgroups) | BIA-T-150204020500-echo-num-tapse-<br>mfas.rtf |
| 72 | Table 15.2.4.3.1 Incidence of Echocardiography Abnormalities – Full Analysis Set | BIA-T-150204030100-echo-abnorm-fas.rtf |
| 73 | Table 15.2.4.3.2 Incidence of Echocardiography Abnormalities – Modified Full Analysis Set | BIA-T-150204030200-echo-abnorm-<br>mfas.rtf |
| 74 | Table 15.2.4.4.1 Shift Table of Echocardiography Results – Full Analysis Set | BIA-T-150204040100-echo-shift-fas.rtf |
| 75 | Table 15.2.4.4.2 Shift Table of Echocardiography Results – Modified Full Analysis Set | BIA-T-150204040200-echo-shift-mfas.rtf |
| 76 | Table 15.2.5.1.1 Summary of NYHA/WHO Functional Class – Full Analysis Set | BIA-T-150205010100-whofc-fas.rtf |
| 77 | Table 15.2.5.1.2 Summary of NYHA/WHO Functional Class – Modified Full Analysis Set | BIA-T-150205010200-whofc-mfas.rtf |
| 78 | Table 15.2.5.2.1 Shift Table of NYHA/WHO Functional Class – Full Analysis Set | BIA-T-150205020100-whofc-shift-fas.rtf |
| 79 | Table 15.2.5.2.2 Shift Table of NYHA/WHO Functional Class – Modified Full Analysis Set | BIA-T-150205020200-whofc-shift-mfas.rtf |
| 80 | Table 15.2.6.1.1 Summary of SF-36v2 Domain Scores by HTD – Full Analysis Set | BIA-T-150206010100-sf36-htd-fas.rtf |
| 81 | Table 15.2.6.1.2 Summary of SF-36v2 Domain Scores – Full Analysis Set | BIA-T-150206010200-sf36-tot-fas.rtf |
| 82 | Table 15.2.6.1.3 Summary of SF-36v2 Domain Scores<br>by HTD – Modified Full Analysis Set | BIA-T-150206010300-sf36-htd-mfas.rtf |
| 83 | Table 15.2.6.1.4 Summary of SF-36v2 Domain Scores – Modified Full Analysis Set | BIA-T-150206010400-sf36-tot-mfas.rtf |
| 84 | Table 15.2.6.2.1 Summary of Norm-Based SF-36v2<br>Scores by HTD – Full Analysis Set | BIA-T-150206020100-sf36-norm-htd-fas.rtf |
| 85 | Table 15.2.6.2.2 Summary of Norm-Based SF-36v2<br>Scores – Full Analysis Set | BIA-T-150206020200-sf36-norm-tot-fas.rtf |
| 86 | Table 15.2.6.2.3 Summary of Norm-Based SF-36v2 Domain Scores by HTD – Modified Full Analysis Set | BIA-T-150206020300-sf36-norm-htd-mfas.rtf |
| 87 | Table 15.2.6.2.4 Summary of Norm-Based SF-36v2 Domain Scores – Modified Full Analysis Set | BIA-T-150206020400-sf36-norm-tot-<br>mfas.rtf |

I-DM-011SAP 

| 88 | Table 15.2.6.3.1 Summary of SF-36v2 Utility Index Scores by HTD – Full Analysis Set | BIA-T-150206030100-sf36-util-htd-fas.rtf |
|---|---|---|
| 89 | Table 15.2.6.3.2 Summary of SF-36v2 Utility Index Scores – Full Analysis Set | BIA-T-150206030200-sf36-util-tot-fas.rtf |
| 90 | Table 15.2.6.3.3 Summary of SF-36v2 Utility Index<br>Scores by HTD – Modified Full Analysis Set | BIA-T-150206030300-sf36-util-htd-mfas.rtf |
| 91 | Table 15.2.6.3.4 Summary of SF-36v2 Utility Index<br>Scores – Modified Full Analysis Set | BIA-T-150206030400-sf36-util-tot-mfas.rtf |
| 92 | Table 15.2.6.4.1 Summary of SF-36v2 Cardio<br>Benchmark Interpretation – Full Analysis Set | BIA-T-150206040100-sf36-cardio-fas.rtf |
| 93 | Table 15.2.6.4.2 Summary of SF-36v2 Cardio Benchmark Interpretation – Modified Full Analysis Set | BIA-T-150206040200-sf36-cardio-mfas.rtf |
| 94 | Table 15.2.6.5.1 Shift Table of SF-36v2 Cardio Benchmark Interpretation – Full Analysis Set | BIA-T-150206050100-sf36-cardio-shift-fas.rtf |
| 95 | Table 15.2.6.5.2 Shift Table of SF-36v2 Cardio Benchmark Interpretation – Modified Full Analysis Set | BIA-T-150206050200-sf36-cardio-shift-<br>mfas.rtf |
| Safet | y Data | |
| 96 | Table 15.3.1.1 Overall Summary of TEAEs – Safety Set | BIA-T-150301010000-teae-sum-ss.rtf |
| 97 | Table 15.3.1.2 Incidence of TEAEs – Safety Set | BIA-T-150301020000-teae-ss.rtf |
| 98 | Table 15.3.1.3 Incidence of Serious TEAEs – Safety Set | BIA-T-150301030000-tesae-ss.rtf |
| 99 | Table 15.3.1.4 Incidence of TEAEs of Special Interest – Safety Set | BIA-T-150301040000-teae-si-ss.rtf |
| 100 | Table 15.3.1.5 Incidence of Related TEAEs – Safety Set | BIA-T-150301050000-teae-rel-ss.rtf |
| 101 | Table 15.3.1.6 Incidence of Related Serious TEAEs – Safety Set | BIA-T-150301060000-tesae-rel-ss.rtf |
| 102 | Table 15.3.1.7 Incidence of TEAEs Leading to Down-<br>Titration – Safety Set | BIA-T-150301070000-teae-dt-ss.rtf |
| 103 | Table 15.3.1.8 Incidence of TEAEs Leading to Discontinuation – Safety Set | BIA-T-150301080000-teae-disc-ss.rtf |
| 104 | Table 15.3.1.9 Incidence of TEAEs Leading to Death – Safety Set | BIA-T-150301090000-teae-death-ss.rtf |
| 105 | Table 15.3.1.10 Incidence of TEAEs by Severity – Safety Set | BIA-T-150301100000-teae-bysev-ss.rtf |
| 106 | Table 15.3.1.11 Incidence of TEAEs by Relationship to IMP – Safety Set | BIA-T-150301110000-teae-byrel-ss.rtf |
| 107 | Table 15.3.2.1.1.1 Summary of Clinical Laboratory Tests: Haematology by HTD– Safety Set | BIA-T-150302010101-lbh-htd-ss.rtf |
| 108 | Table 15.3.2.1.1.2 Summary of Clinical Laboratory Tests: Haematology– Safety Set | BIA-T-150302010102-lbh-tot-ss.rtf |
| 109 | Table 15.3.2.1.2.1 Summary of Clinical Laboratory Tests: Biochemistry by HTD – Safety Set | BIA-T-150302010201-lbb-htd-ss.rtf |
| 110 | Table 15.3.2.1.2.2 Summary of Clinical Laboratory Tests: Biochemistry – Safety Set | BIA-T-150302010202-lbb-tot-ss.rtf |
| 111 | SetTable 15.3.2.1.3.1 Summary of Clinical Laboratory<br>Tests: Coagulation by HTD – Safety Set | BIA-T-150302010301-lbco-htd-ss.rtf |
| 112 | Table 15.3.2.1.3.2 Summary of Clinical Laboratory Tests: Coagulation – Safety Set | BIA-T-150302010302-lbco-tot-ss.rtf |
| 113 | Table 15.3.2.1.4 Summary of Clinical Laboratory Tests: Urinalysis – Safety Set | BIA-T-150302010400-lbu-ss.rtf |
| 114 | Table 15.3.2.2.1 Clinical Laboratory Tests: Incidence of Haematology Abnormalities – Safety Set | BIA-T-150302020100-lbh-abnorm-ss.rtf |
| 115 | Table 15.3.2.2.2 Clinical Laboratory Tests: Incidence of Biochemistry Abnormalities – Safety Set | BIA-T-150302020200-lbb-abnorm-ss.rtf |
| 116 | Table 15.3.2.2.3 Clinical Laboratory Tests: Incidence of Coagulation Abnormalities – Safety Set | BIA-T-150302020300-lbco-abnorm-ss.rtf |
| 117 | Table 15.3.2.2.4 Clinical Laboratory Tests: Incidence of Urinalysis Abnormalities – Safety Set | BIA-T-150302020400-lbu-abnorm-ss.rtf |
| 118 | Table 15.3.2.3.1 Clinical Laboratory Tests: Shift Table of Haematology Results – Safety Set | BIA-T-150302030100-lbh-shift-ss.rtf |
| 119 | Table 15.3.2.3.2 Clinical Laboratory Tests: Shift Table | BIA-T-150302030200-lbb-shift-ss.rtf |

I-DM-011SAP 

| 120 | Table 15.3.2.3.3 Clinical Laboratory Tests: Shift Table | BIA-T-150302030300-lbco-shift-ss.rtf |
|---|---|---|
| | of Coagulation Results – Safety Set | |
| 121 | Table 15.3.2.3.4 Clinical Laboratory Tests: Shift Table | BIA-T-150302030400-lbu-shift-ss.rtf |
| | of Urinalysis Results – Safety Set | |
| 122 | Table 15.3.3.1.1 Summary of Arterial Blood Gas | BIA-T-150303010100-artbg-htd-ss.rtf |
| | Analysis by HTD– Safety Set | |
| 123 | Table 15.3.3.1.2 Summary of Arterial Blood Gas | BIA-T-150303010200-artbg-tot-ss.rtf |
| | Analysis – Safety Set | |
| 124 | Table 15.3.3.2 Incidence of Arterial Blood Gas | BIA-T-150303020000-artbg-abnorm-ss.rtf |
| | Analysis Abnormalities – Safety Set | |
| 125 | Table 15.3.3.3 Shift Table of Arterial Blood Gas | BIA-T-150303030000-artbg-shift-ss.rtf |
| | Analysis Results – Safety Set | |
| 126 | Table 15.3.3.4.1 Summary of Peripheral Oxygen | BIA-T-150303040100-po2-htd-ss.rtf |
| | Saturation (%) by HTD– Safety Set | 1 |
| 127 | Table 15.3.3.4.2 Summary of Peripheral Oxygen | BIA-T-150303040200-po2-tot-ss.rtf |
| 127 | Saturation (%) – Safety Set | Bir 1 1303030 10200 po2 tot ss.iti |
| 128 | Table 15.3.4.1.1 Summary of Vital Signs by HTD – | BIA-T-150304010100-vs-htd-ss.rtf |
| 120 | Safety Set | B11-1-13030-010100-v3-11tt-35.1tt |
| 129 | Table 15.3.4.1.2 Summary of Vital Signs – Safety Set | BIA-T-150304010200-vs-tot-ss.rtf |
| 130 | Table 15.3.4.2 Summary of Vital Signs by Pooled | BIA-T-150304020000-vs-htdpool-ss.rtf |
| | HTD – Safety Set | |
| 131 | Table 15.3.4.3.1 Summary of Short-Term IMP Effect | BIA-T-150304030100-vs-visitchg-htd-ss.rtf |
| | on Vital Signs by HTD – Safety Set | |
| 132 | Table 15.3.4.3.2 Summary of Short-Term IMP Effect | BIA-T-150304030200-vs-visitchg-tot-ss.rtf |
| | on Vital Signs – Safety Set | |
| 133 | Table 15.3.4.4.1 Summary of Change in Short-Term | BIA-T-150304040100-vs-effchg-htd-ss.rtf |
| | IMP Effect on Vital Signs by HTD – Safety Set | <i>g</i> |
| 134 | Table 15.3.4.4.2 Summary of Change in Short-Term | BIA-T-150304040200-vs-effchg-tot-ss.rtf |
| | IMP Effect on Vital Signs – Safety Set | |
| 135 | Table 15.3.4.5.1 Summary of Physical Measurements | BIA-T-150304050100-physmeas-htd-ss.rtf |
| 133 | by HTD – Safety Set | Birr i 13030 1030100 pirysineds file ss.iti |
| 136 | Table 15.3.4.5.2 Summary of Physical Measurements – | BIA-T-150304050200-physmeas-tot-ss.rtf |
| 130 | Safety Set | B11-1-130304030200-pitysineas-tot-ss.iti |
| 137 | Table 15.3.5.1.1 Summary of ECG Assessments by | BIA-T-150305010100-ecg-htd-ss.rtf |
| 137 | HTD – Safety Set | BIA-1-130303010100-ccg-litt-ss.iti |
| 138 | Table 15.3.5.1.2 Summary of ECG Assessments – | BIA-T-150305010200-ecg-tot-ss.rtf |
| 130 | Safety Set | BIA-1-130303010200-ccg-tot-ss.tti |
| 139 | Table 15.3.5.2.1 Summary of Short-Term IMP Effect | BIA-T-150305020100-ecg-visitchg-htd- |
| 139 | | ss.rtf |
| 1.40 | on ECG Assessments by HTD – Safety Set | |
| 140 | Table 15.3.5.2.2 Summary of Short-Term IMP Effect | BIA-T-150305020200-ecg-visitchg-tot- |
| 1 / 1 | on ECG Assessments – Safety Set | ss.rtf |
| 141 | Table 15.3.5.3.1 Summary of Change in Short-Term | BIA-T-150305030100-ecg-effchg-htd-ss.rtf |
| | IMP Effect on ECG Assessements by HTD – Safety | |
| 1.42 | Set | DIA T 150205020200 CC1 |
| 142 | Table 15.3.5.3.2 Summary of Change in Short-Term | BIA-T-150305030200-ecg-effchg-tot-ss.rtf |
| | IMP Effect on ECG Assessements – Safety Set | DV. 7.470207040405 |
| 143 | Table 15.3.5.4.1 Incidence of ECG Abnormalities – | BIA-T-150305040100-ecg-abnorm-ss.rtf |
| | Safety Set | |
| 144 | Table 15.3.5.4.2 Shift Table of ECG Abnormalities – | BIA-T-150305040200-ecg-shift-ss.rtf |
| | Safety Set | |
| 145 | Table 15.3.5.4.3 Shift Table of Within-Visit ECG | BIA-T-150305040300-ecg-shift-visit-ss.rtf |
| | Abnormalities – Safety Set | |
| 146 | Table 15.3.6 Summary of Physical Examination | BIA-T-150306000000-pe-ss.rtf |
| | Findings – Safety Set | |
| 147 | Table 15.3.7.1 Summary of Scleroderma Scarring by | BIA-T-150307010000-sclero-htd-ss.rtf |
| | HTD – Safety Set | |
| 148 | Table 15.3.7.2 Summary of Scleroderma Scarring – | BIA-T-150307020000-sclero-tot-ss.rtf |
| 1.0 | Safety Set | |
| 149 | Table 15.3.8.1 Summary of mRSS by HTD – Safety | BIA-T-150308010000-mrss-htd-ss.rtf |
| 17/ | Set | 211 1 10000010000-mmss-mu-ss.m |
| 150 | Table 15.3.8.2 Summary of mRSS – Safety Set | BIA-T-150308020000-mrss-tot-ss.rtf |
| 150 | 14010 13.3.0.2 Summary of mixes – Safety Set | D11 - 1 - 1 50 50 00 20 000 - HH 55 - 10 1 - 55 . HI |

I-DM-011SAP 

# 10.2 Listings

Appendix listings defined below will be provided to the sponsor in separate .rtf files for each output.

| No | Listing Identifier, Title | Output file |
|---|---|---|
| Dem | Demographic and Study Population Data | |
| 1 | Listing 16.2.1.1.1 Patient Disposition – Safety Set | BIA-L-1602010101-disp-ss.rtf |
| 2 | Listing 16.2.1.1.2 Screening Failures – Enrolled Set | BIA-L-1602010102-scrfail-enr.rtf |
| 3 | Listing 16.2.1.2 Patient Visits – Enrolled Set | BIA-L-1602010200-visits-enr.rtf |
| 4 | Listing 16.2.1.3.1 Major Protocol Deviations – Safety Set | BIA-L-1602010301-protdev-ss.rtf |
| 5 | Listing 16.2.1.3.2 Patients Affected by the COVID-19 Pandemic – Safety Set | BIA-L-1602010302-protdev-covid-ss.rtf |
| 6 | Listing 16.2.1.3.3 Inclusion Criteria Not Met and Exclusion Criteria Met – Enrolled Set | BIA-L-1602010303-ie-enr.rtf |
| 7 | Listing 16.2.1.4 Exclusions from Analysis Sets –<br>Enrolled Set | BIA-L-1602010400-anlset-excl-enr.rtf |
| 8 | Listing 16.2.1.5 Demographics and Baseline<br>Characteristics – Enrolled Set | BIA-L-1602010500-demo-enr.rtf |
| 9 | Listing 16.2.1.6 Disease Characteristics – Enrolled Set | BIA-L-1602010600-diseasechar-enr.rtf |
| 10 | Listing 16.2.1.7 Medical History – Enrolled Set | BIA-L-1602010700-mh-enr.rtf |
| 11 | Listing 16.2.1.8 Medications and Therapies – Enrolled Set | BIA-L-1602010800-conmed-enr.rtf |
| 12 | Listing 16.2.2.1 Drug Accountability- Safety Set | BIA-L-1602020100-da-ss.rtf |
| 13 | Listing 16.2.2.2 Exposure to IMP and Compliance – Safety Set | BIA-L-1602020200-imp-compl-ss.rtf |
| Effic | acy Data | |
| 14 | Listing 16.2.3.1 Right Heart Catheterization Parameters – Enrolled Set | BIA-L-1602030100-rhc-enr.rtf |
| 15 | Listing 16.2.3.2 6-Min Walking Test – Enrolled Set | BIA-L-1602030200-6mwt-enr.rtf |
| 16 | Listing 16.2.3.3 Biomarker NT-proBNP – Enrolled Set | BIA-L-1602030300-biomarker-enr.rtf |
| 17 | Listing 16.2.3.4 Echocardiography – Enrolled Set | BIA-L-1602030400-echo-enr.rtf |
| 18 | Listing 16.2.3.5 NYHA/WHO Functional Class – Enrolled Set | BIA-L-1602030500-whofe-enr.rtf |
| 19 | Listing 16.2.3.6 SF-36v2 – Enrolled Set | BIA-L-1602030600-sf36-enr.rtf |
| Safet | y Data | |
| 20 | Listing 16.2.4.1.1 Adverse Events: MedDRA Coding | BIA-L-1602040101-aecod.rtf |
| 21 | Listing 16.2.4.1.2 Adverse Events: General – Enrolled Set | BIA-L-1602040102-ae-enr.rtf |
| 22 | Listing 16.2.4.1.3 Non-Serious Adverse Events – Safety Set | BIA-L-1602040103-nsae-ss.rtf |
| 23 | Listing 16.2.4.1.4 Serious Adverse Events – Safety Set | BIA-L-1602040104-sae-ss.rtf |
| 24 | Listing 16.2.4.1.5 TEAEs of Special Interest - Safety Set | BIA-L-1602040105-teae-si-ss.rtf |
| 25 | Listing 16.2.4.1.6 AEs Leading to Discontinuation – Safety Set | BIA-L-1602040106-ae-disc-ss.rtf |
| 26 | Listing 16.2.4.1.7 AEs Leading to Death – Safety Set | BIA-L-1602040107-ae-death-ss.rtf |
| 27 | Listing 16.2.4.2.1 Laboratory Data: Haematology – Enrolled Set | BIA-L-1602040201-lbh-enr.rtf |
| 28 | Listing 16.2.4.2.2 Laboratory Data: Biochemistry – Enrolled Set | BIA-L-1602040202-lbb-enr.rtf |
| 29 | Listing 16.2.4.2.3 Laboratory Data: Coagulation – Enrolled Set | BIA-L-1602040203-lbco-enr.rtf |
| 30 | Listing 16.2.4.2.4 Laboratory Data: Urinalysis – Enrolled Set | BIA-L-1602040204-lbu-enr.rtf |

I-DM-011SAP 

| 31 | Listing 16.2.4.2.5 Laboratory Data: Microscopy – | BIA-L-1602040205-lbmicro-enr.rtf |
|---|---|---|
| | Enrolled Set | |
| 32 | Listing 16.2.4.2.6 Laboratory Data: Pregnancy Tests – | BIA-L-1602040206-lbpreg-enr.rtf |
| | Enrolled Set | |
| 33 | Listing 16.2.4.3 Arterial Blood Gas Analysis – | BIA-L-1602040300-artbg-enr.rtf |
| | Enrolled Set | |
| 34 | Listing 16.2.4.4 Vital Signs – Enrolled Set | BIA-L-1602040400-vs-enr.rtf |
| 35 | Listing 16.2.4.5 Electrocardiogram – Enrolled Set | BIA-L-1602040500-ecg-enr.rtf |
| 36 | Listing 16.2.4.6 Physical Examinations – Enrolled Set | BIA-L-1602040600-pe-enr.rtf |
| 37 | Listing 16.2.4.7 Number of Digital Scars – Enrolled | BIA-L-1602040700-scars-enr.rtf |
| | Set | |
| 38 | Listing 16.2.4.8 Modified Rodnan Skin Score – | BIA-L-1602040800-mrss-enr.rtf |
| | Enrolled Set | |

I-DM-011SAP Effective date: 15.09.2020 

# 10.3 Figures

Appendix figures defined below will be provided to the sponsor in separate .rtf files for each output.

| No | Figure Identifier, Title | Output file |
|---|---|---|
| Dem | ographic and Study Population Data | |
| 1 | Figure 15.1.1 Flow Chart of Patient Disposition – Enrolled Set | BIA-F-15010100-disp-enr.rtf |
| 2 | Figure 15.1.2 Flow Chart of Analysis Sets – Enrolled Set | BIA-F-15010200-anlset-enr.rtf |
| Effic | acy Data | |
| 3 | Figure 15.2.1.1 Box-Whisker Plot of NT-proBNP by Pooled HTD – Full Analysis Set | BIA-F-15020101-biomarker-htdpool-<br>fas.rtf |
| 4 | Figure 15.2.1.2 Box-Whisker Plot of NT-proBNP by Pooled HTD – Modified Full Analysis Set | BIA-F-15020102-biomarker-htdpool-<br>mfas.rtf |
| 5 | Figure 15.2.2.1 Norm-Based SF-36v2 Domain Scores by Visit – Full Analysis Set | BIA-F-15020201-sf36-norm-fas.rtf |
| 6 | Figure 15.2.2.2 Norm-Based SF-36v2 Domain Scores by Visit – Modified Full Analysis Set | BIA-F-15020202-sf36-norm-mfas.rtf |
| 7 | Figure 15.2.3.1 SF-36v2 Cardio Benchmark Interpretation by<br>Visit – Full Analysis Set | BIA-F-15020301-sf36-cardio-fas.rtf |
| 8 | Figure 15.2.3.2 SF-36v2 Cardio Benchmark Interpretation by Visit – Modified Full Analysis Set | BIA-F-15020302-sf36-cardio-mfas.rtf |
| Safe | ty Data | |
| 9 | Figure 15.3.1 Vital Signs Median Change from Baseline – Safety Set | BIA-F-15030100-vs-med-ss.rtf |

I-DM-011SAP 

# **SIGNATURES**

| Signature Author: Lukas Pukys Statistician, Scope International AG Vilnius, Lithuania | Date |
|---|---|
| Signature Reviewer: Giedrius Vilutis Statistician, Scope International AG Vilnius, Lithuania | |
| Signature<br>Sponsor:<br>Ana Santos<br>Clinical Operations Manager (\$OC2), I<br>Coronado, Portugal | <i>Date</i> Bial - Portela & C <sup>a</sup> , S.A. |
| Signature<br>Sponsor:<br>Luís Magalhães<br>Head of Clinical Research, Bial - Porte<br>Coronado, Portugal | Date |
| Signature<br>Sponsor:<br>Guillermo Castilla<br>Biostatistician, Bial - Portela & C <sup>a</sup> , S.A<br>Coronado, Portugal | Date |

I-DM-011SAP Effective date: 15.09.2020 